CLINICAL TRIAL: NCT00833989
Title: A Single-Blind Study of the Safety, Pharmacokinetics and Pharmacodynamics of Escalating Repeat Doses of GSK249320 in Patients With Stroke
Brief Title: Safety Escalating Repeat IV, in Stroke Patients
Acronym: MAG111539
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 111539
Record Dates: First submitted 2009-01-29; First posted 2009-02-02 (Estimated); Results first posted 2017-10-16 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-09

CONDITIONS: Ischaemic Attack, Transient
MeSH Terms: interventions — refanezumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- PLACEBO (Placebo Comparator)
  Interventions: Drug: PLACEBO
- ACTIVE (Experimental)
  Interventions: Drug: GSK249320

INTERVENTIONS:
Drug: GSK249320 — I.V. infusion
  Arms: ACTIVE
Drug: PLACEBO — Placebo
  Arms: PLACEBO

SUMMARY:
The purpose of this study is to is to test increasing repeat doses of GSK249320 compared to placebo in patients with stroke.

DETAILED DESCRIPTION:
GSK249320 is a humanised monoclonal antibody (mAb) that binds with high specificity to myelin-associated glycoprotein (MAG) and antagonises or neutralises MAG-mediated inhibition and has been shown to improve functional recovery after stroke in pre-clinical models, possibly by promoting neuroregeneration and plasticity. The present study is the first in patients with stroke. The main aim of this study is to select tolerated doses of GSK249320 that can be used in future trials to evaluate its efficacy in improving clinical function in patients recovering from stroke. This clinical trial is designed as a placebo-controlled, single-blind, multicenter study to investigate the safety, pharmacokinetics (PK) and pharmacodynamics (PD) of escalating repeat IV doses of GSK249320. Three sequential dose escalation cohorts (1, 5 and 15 mg/kg) are planned, with 8 patients on placebo and 8 on active in cohort 1 and 4 patients on placebo and 8 on active in cohorts 2 and 3. Each patient will receive 2 repeat IV doses 9 ± 1 days apart and assessments will extend to at least 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed diagnosis of stroke
* Stroke onset must be within the last 24-72 hours.
* Have a stroke that is either:
* radiologically confirmed to be ischaemic and supratentorial. The diameter of the ischemic lesion is >15mm in any singlle direction or the volume is >4cc. OR
* radiologically confirmed to be an intracerebral hemorrhage that is supratentorial, deep (i.e., blood must not directly contact cerebral cortex) and with minimal or no intraventricular extension. The Intracerebral Hemorrahage (CH) score must be 0-2 and is calculated based on age, Galsgow coma Scale score ad the initial CT or MRI findings for the index stroke. See the SOM for the full calculation procedure.
* Have a total NIHSS score of 3-21.
* Have an upper and/or lower limb deficit defined as:
* Score of 1-3 on the NIHSS Motor Arm question, and palpable and observable voluntary extension or flexion of the fingers. AND/OR b. Score of 1-3 on the NIHSS Motor Leg question
* Aged 18-90, inclusive.
* Male subjects and females of non-child-bearing potential are allowed to participate in this study.
* Females of child-bearing potential are also allowed to participate in this study provided they are using a contraceptive method with a failure rate of <1%.

Exclusion Criteria:

* History of a previous symptomatic stroke within 3 months prior to study entry.
* Presence of significant disability prior to the current stroke. Significant disability is defined as having a pre-stroke Rankin score of >2.
* Presence of depression that is active and not adequately controlled such that it interferred with major activities of daily living immediately prior to the current stroke.
* Subjects who are not alert or are unresponsive as defined by a score of 2 or 3 on the NIHSS Level of Consciousness question (question #1a).
* Presence of significant aphasia as likely to confound or interfere with completion of the study assessments.
* Presence of peripheral neuropathy, including diabetic neuropathy, which is clinically active and symptomatic at time of screening.
* Presence of neurological or psychiatric disease, such as dementia or mild cognitive impairment, prior to study entry that is likely to confound clinical evaluations.
* Presence of a demyelinating disease, such as multiple sclerosis.
* Evidence of other chronic co-morbid conditions or unstable acute systemic illnesses which, in the opinion of the investigator, could shorten the subject's survival or limit his/her ability to complete the study.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Presence of QTcB > 500 msec; or uncorrected QT >600msec (machine or manual over-read) on baseline ECG.
* Contraindication to TMS, such as:
* have metal present, such as hardware or plate on the scalp in the area to which TMS will be applied, implanted cardiac pacemaker, implanted prosthetic heart valve, medication pump or line, metallic implant or clip in the head/neck, electrical, mechanical or magnetic implants, neuro-stimulation device, or orthodontic work involving ferromagnetic materials
* occupation or activity that may cause accidental lodging of ferromagnetic materials or embedded metal fragments in the head. Subjects can be cleared by a head computed tomography scan.
* concomitant use of drugs that substantially lower seizure threshold (e.g., tricyclic antidepressants and neuroleptics)
* known history of seizures or epilepsy
* brain tumor, recent brain injury (within 5 years) associated with definite loss of consciousness, or any history of brain surgery
* Contraindication to MRI, such as:
* have metal present, such as implanted cardiac pacemaker, implanted prosthetic heart valve, medication pump or line, metallic implant or clip in the head/neck, electrical, mechanical or magnetic implants, neuro-stimulation device, or orthodontic work involving ferromagnetic materials, permanent tattooed metallic eye-liner
* occupation or activity that may cause accidental lodging of ferromagnetic materials or embedded metal fragments in the head. Subjects can be cleared by a head computed tomography scan.
* claustrophobia
* Participation in any investigational rehabilitation paradigm targeting stroke recovery during the duration of this study.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).

Pregnant or lactating females.

* Subjects considered unwilling or unable to comply with the procedures and study visit schedule outlined in the protocol.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-07-08 (Actual); Primary Completion 2011-01-31 (Actual); Study Completion 2011-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- United States (5):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Fort Collins, Colorado
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Portland, Oregon
- Canada (2):
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- Germany (8):
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Celle, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Leipzig, Saxony

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Cramer SC, Abila B, Scott NE, Simeoni M, Enney LA; MAG111539 Study Investigators. Safety, pharmacokinetics, and pharmacodynamics of escalating repeat doses of GSK249320 in patients with stroke. Stroke. 2013 May;44(5):1337-42. doi: 10.1161/STROKEAHA.111.674366. Epub 2013 Mar 7. PMID 23471268
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 111539 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111539 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111539 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111539 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111539 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111539 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111539 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 08-July-2009 and 31-January-2011 at 15 centers in 3 countries including 2 centers in Canada, 8 centers in Germany and 5 centers in the United States. Of the 15 centers, 10 centers enrolled participants.
Pre-assignment Details: A total of 42 participants were randomized and included in All subject population.
Groups:
- Placebo: Eligible participants received 0.9% Sodium chloride as an intravenous (IV) infusion via a programmable infusion pump. Each participant received two IV doses 9 ±1 days apart, where the first dose was administered 24-72 hours post stroke. Assessments for safety, pharmacokinetics and pharmacodynamics markers were extended to at least 16 weeks.
- GSK249320 1 mg/kg: Eligible participants received GSK249320, 1 milligram per kilogram (mg/kg)of body weight as an IV infusion via a programmable infusion pump. Each participant received two IV doses 9 ±1 days apart, where the first dose was administered 24-72 hours post stroke. Assessments for safety, pharmacokinetics and pharmacodynamics markers were extended to at least 16 weeks.
- GSK249320 5 mg/kg: Eligible participants received GSK249320, 5mg/kg of body weight as an IV infusion via a programmable infusion pump. Each participant received two IV doses 9 ±1 days apart, where the first dose was administered 24-72 hours post stroke. Assessments for safety, pharmacokinetics and pharmacodynamics markers were extended to at least 16 weeks.
- GSK249320 15 mg/kg: Eligible participants received GSK249320, 15mg/kg of body weight as an IV infusion via a programmable infusion pump. Each participant received two IV doses 9 ±1 days apart, where the first dose was administered 24-72 hours post stroke. Assessments for safety, pharmacokinetics and pharmacodynamics markers were extended to at least 16 weeks
Period: Overall Study
Arm/Group | Placebo | GSK249320 1 mg/kg | GSK249320 5 mg/kg | GSK249320 15 mg/kg
Started | 17 | 8 | 9 | 8
Completed | 14 | 8 | 8 | 6
Not Completed | 3 | 0 | 1 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Eligible participants received 0.9% Sodium chloride as an IV infusion via a programmable infusion pump. Each participant received two IV doses 9 ±1 days apart, where the first dose was administered 24-72 hours post stroke. Assessments for safety, pharmacokinetics and pharmacodynamics markers were extended to at least 16 weeks.
- GSK249320 1 mg/kg: Eligible participants received GSK249320, 1 mg/kg of body weight as an IV infusion via a programmable infusion pump. Each participant received two IV doses 9 ±1 days apart, where the first dose was administered 24-72 hours post stroke. Assessments for safety, pharmacokinetics and pharmacodynamics markers were extended to at least 16 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK249320 1 mg/kg | GSK249320 5 mg/kg | GSK249320 15 mg/kg | Total
Number analyzed (Participants) | 17 | 8 | 9 | 8 | 42
Age, Continuous [Mean (Standard Deviation); unit: Year] | 67.6 (10.79) | 62.1 (13.01) | 63.9 (13.76) | 59.3 (12.99) | 64.2 (12.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 3 | 5 | 4 | 23
  Male | 6 | 5 | 4 | 4 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 17 | 7 | 9 | 7 | 40
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 00 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: AE was defined as any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE include AEs those result in death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
Time Frame: Up to 112 days
Population: All Subjects population was defined as all participants who receive at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK249320 1 mg/kg | GSK249320 5 mg/kg | GSK249320 15 mg/kg
Number analyzed (Participants) | 17 | 8 | 9 | 8
Participants
  Any AE | 11 | 6 | 8 | 6
  Any SAE | 3 | 1 | 3 | 3

2. Primary Outcome: Number of Participants With Vital Signs Changes of Potential Clinical Importance
Description: The potential clinical importance ranges (low and high) of the vital sign parameters were for systolic blood pressure (SBP) (<85 and >200 millimeter of mercury [mmHg]), diastolic blood pressure (DBP) (<45 and >110 mmHg) and heart rate (HR) (<40 and >110 beats per minute). Only those parameters for which at least one value of potential clinical importance was reported are summarized. The number of participants with potential clinical important vital parameter findings at any visit were reported.
Time Frame: Up to 112 days
Population: All Subjects population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK249320 1 mg/kg | GSK249320 5 mg/kg | GSK249320 15 mg/kg
Number analyzed (Participants) | 17 | 8 | 9 | 8
Participants
  SBP, Visit 1, Day 1, 30 minute, High | 1 | 0 | 0 | 0
  SBP, Visit 1, Day 1, 1 hour, High: number analyzed (Participants) | 16 | 8 | 9 | 7
  SBP, Visit 1, Day 1, 1 hour, High | 1 | 0 | 0 | 0
  SBP, Visit 1, Day 1, 1 hour, Low: number analyzed (Participants) | 16 | 8 | 9 | 7
  SBP, Visit 1, Day 1, 1 hour, Low | 1 | 0 | 0 | 0
  SBP, Visit 1, Day 1, 2 hour, High: number analyzed (Participants) | 17 | 7 | 9 | 8
  SBP, Visit 1, Day 1, 2 hour, High | 2 | 0 | 0 | 0
  SBP, Visit 1, Day 1, 4 hour, High: number analyzed (Participants) | 17 | 7 | 8 | 8
  SBP, Visit 1, Day 1, 4 hour, High | 1 | 0 | 0 | 1
  SBP, Visit 1, Day 1, 8 hour, High: number analyzed (Participants) | 17 | 7 | 9 | 8
  SBP, Visit 1, Day 1, 8 hour, High | 1 | 0 | 0 | 0
  SBP, Visit 1, Day 1, 12 hour, High | 0 | 1 | 0 | 1
  SBP, Visit 1, Day 1, 12 hour, Low | 0 | 0 | 1 | 0
  SBP, Visit 1, Day 1, 24 hour, High: number analyzed (Participants) | 16 | 8 | 9 | 8
  SBP, Visit 1, Day 1, 24 hour, High | 0 | 0 | 1 | 0
  SBP, Visit 6, Day 90, Low: number analyzed (Participants) | 14 | 8 | 8 | 6
  SBP, Visit 6, Day 90, Low | 0 | 0 | 1 | 0
  SBP, Visit 7, Day 112, Low | 1 | 0 | 0 | 0
  DBP, Visit 1, Day 1, 15 minute, Low | 0 | 0 | 1 | 0
  DBP, Visit 1, Day 1, 1 hour, High: number analyzed (Participants) | 16 | 8 | 9 | 7
  DBP, Visit 1, Day 1, 1 hour, High | 1 | 0 | 0 | 0
  DBP, Visit 1, Day 1, 2 hour, High: number analyzed (Participants) | 17 | 7 | 9 | 8
  DBP, Visit 1, Day 1, 2 hour, High | 1 | 0 | 0 | 0
  DBP, Visit 1, Day 1, 2 hour, Low | 0 | 1 | 0 | 0
  DBP, Visit 1, Day 1, 4 hour, High: number analyzed (Participants) | 17 | 7 | 8 | 8
  DBP, Visit 1, Day 1, 4 hour, High | 0 | 1 | 0 | 0
  DBP, Visit 1, Day 1, 12 hour, High | 1 | 0 | 0 | 0
  DBP, Visit 2, Day 5, High: number analyzed (Participants) | 15 | 8 | 9 | 8
  DBP, Visit 2, Day 5, High | 0 | 0 | 1 | 0
  DBP, Visit 3, Day 10, 30 minute, High: number analyzed (Participants) | 14 | 8 | 9 | 7
  DBP, Visit 3, Day 10, 30 minute, High | 1 | 0 | 0 | 0
  HR, Visit 1, Day 1, 0 hour, High | 0 | 1 | 0 | 0
  HR, Visit 1, Day 1, 15 minute, High | 0 | 1 | 0 | 0
  HR, Visit 1, Day 1, 30 minute, High | 1 | 1 | 0 | 0
  HR, Visit 1, Day 1, 45 minute, High: number analyzed (Participants) | 17 | 8 | 9 | 7
  HR, Visit 1, Day 1, 45 minute, High | 1 | 1 | 1 | 0
  HR, Visit 1, Day 1, 1 hour, High: number analyzed (Participants) | 16 | 8 | 9 | 6
  HR, Visit 1, Day 1, 1 hour, High | 0 | 1 | 0 | 0
  HR, Visit 1, Day 1, 2 hour, High: number analyzed (Participants) | 17 | 7 | 9 | 8
  HR, Visit 1, Day 1, 2 hour, High | 0 | 1 | 1 | 0
  HR, Visit 1, Day 1, 12 hour, High | 0 | 0 | 1 | 0
  HR, Visit 1, Day 1, 24 hour, High: number analyzed (Participants) | 16 | 8 | 9 | 8
  HR, Visit 1, Day 1, 24 hour, High | 0 | 0 | 0 | 1
  HR, Visit 2, Day 5, High: number analyzed (Participants) | 15 | 8 | 9 | 8
  HR, Visit 2, Day 5, High | 0 | 0 | 1 | 0
  HR, Visit 3, Day 10, 0 hour, High: number analyzed (Participants) | 14 | 8 | 9 | 7
  HR, Visit 3, Day 10, 0 hour, High | 1 | 1 | 0 | 0
  HR, Visit 3, Day 10, 15 minute, High: number analyzed (Participants) | 14 | 8 | 9 | 7
  HR, Visit 3, Day 10, 15 minute, High | 0 | 1 | 0 | 0
  HR, Visit 3, Day 10, 30 minute, High: number analyzed (Participants) | 14 | 8 | 9 | 7
  HR, Visit 3, Day 10, 30 minute, High | 1 | 1 | 0 | 0
  HR, Visit 3, Day 10, 45 minute, High: number analyzed (Participants) | 14 | 8 | 9 | 7
  HR, Visit 3, Day 10, 45 minute, High | 1 | 1 | 0 | 0
  HR, Visit 3, Day 10, 1 hour, High: number analyzed (Participants) | 14 | 8 | 9 | 7
  HR, Visit 3, Day 10, 1 hour, High | 1 | 0 | 0 | 0
  HR, Visit 3, Day 10, 3 hour, High: number analyzed (Participants) | 14 | 7 | 9 | 7
  HR, Visit 3, Day 10, 3 hour, High | 1 | 0 | 0 | 0
  HR, Visit 4, Day 30, High: number analyzed (Participants) | 14 | 8 | 9 | 7
  HR, Visit 4, Day 30, High | 0 | 1 | 0 | 0

3. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Values Outside Range of Potential Clinical Importance
Description: Single 12-lead ECGs was obtained. The standard ECG criteria of potential clinical importance were uncorrected QT interval <300 and >600 milliseconds (msec), absolute QTc interval >500 msec, increase from Baseline QTc >60 msec, RR Interval <90 and >2000 msec, PR Interval <110 and >220 msec, QRS Interval <75 and >110 msec. The number of participants with potentially clinically significant ECG abnormality were reported.
Time Frame: Up to 112 days
Population: All Subjects population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK249320 1 mg/kg | GSK249320 5 mg/kg | GSK249320 15 mg/kg
Number analyzed (Participants) | 17 | 8 | 9 | 8
Participants
  Visit 1, Day 1, Predose | 2 | 1 | 1 | 0
  Visit 1, Day 1, 24 hour: number analyzed (Participants) | 15 | 7 | 8 | 8
  Visit 1, Day 1, 24 hour | 2 | 1 | 1 | 0
  Visit 2, Day 5: number analyzed (Participants) | 14 | 8 | 9 | 8
  Visit 2, Day 5 | 2 | 0 | 0 | 0
  Visit 3, Day 10, Predose: number analyzed (Participants) | 14 | 7 | 9 | 7
  Visit 3, Day 10, Predose | 2 | 0 | 1 | 0
  Visit 3, Day 10, 3 hour: number analyzed (Participants) | 13 | 7 | 8 | 7
  Visit 3, Day 10, 3 hour | 2 | 1 | 1 | 0
  Visit 4, Day 30: number analyzed (Participants) | 14 | 8 | 9 | 7
  Visit 4, Day 30 | 1 | 1 | 1 | 0
  Visit 5, Day 60: number analyzed (Participants) | 14 | 7 | 9 | 7
  Visit 5, Day 60 | 1 | 0 | 1 | 0
  Visit 6, Day 90: number analyzed (Participants) | 14 | 8 | 8 | 6
  Visit 6, Day 90 | 1 | 0 | 0 | 0
  Visit 7, Day 112: number analyzed (Participants) | 14 | 8 | 6 | 6
  Visit 7, Day 112 | 1 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Nerve Conduction Testing (NCT) Values
Description: NCT (electrode placement technique) of sensory and motor function was performed on the unaffected side (i.e., side that is not affected by the stroke) by appropriately qualified personnel at specified visits (Day 5 and 30 and at early withdrawal). Qualified technician performed the testing; however the same neurologist interpreted the NCT data within a single participant. Both upper and lower extremity nerves were tested and the data was recorded. Number of participants with normal and abnormal NCT data were reported.
Time Frame: Day 5 and 30 and at early withdrawal
Population: All Subject population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK249320 1 mg/kg | GSK249320 5 mg/kg | GSK249320 15 mg/kg
Number analyzed (Participants) | 17 | 8 | 9 | 8
Participants
  Motor, Visit 2, Day 5, Normal | 11 | 7 | 7 | 4
  Motor, Visit 2, Day 5, Abnormal, secondary to | 4 | 1 | 2 | 4
  Motor, Visit 4, Day 30, Normal | 11 | 7 | 6 | 4
  Motor, Visit 4, Day 30, Abnormal, secondary to | 3 | 1 | 2 | 3
  Motor, Early Withdrawal, Abnormal, secondary to | 2 | 0 | 0 | 0
  Sensory, Visit 2, Day 5, Normal | 9 | 4 | 6 | 3
  Sensory, Visit 2, Day 5, Abnormal, secondary to | 5 | 4 | 3 | 5
  Sensory, Not done | 1 | 0 | 0 | 0
  Sensory, Visit 4, Day 30, Normal | 12 | 5 | 7 | 3
  Sensory, Visit 4, Day 30, Abnormal, secondary to | 2 | 3 | 1 | 4
  Sensory, Early Withdrawal, Normal, | 1 | 0 | 0 | 0
  Sensory, Early Withdrawal, Abnormal, secondary to | 1 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With White Matter Changes and Demyelination Assessed by Magnetic Resonance Imaging (MRI)
Description: Whole brain MRI scans were performed by appropriately qualified personnel at those specified visits (Day 1, 10 and 60 or at early withdrawal [if participant withdrew from study before Day 60 MRI]). Required pulse sequences of diffusion weighted imaging (DWI), T1, and T2 FLAIR was performed to measure lesion volume and to look for the presence of any new acute inflammatory lesions. The investigator or other medically qualified study team member evaluated the Day 10 and 60 scans for any new abnormalities or clinically significant worsening. Digital data for each MRI was sent to a central MRI laboratory for an over-read of the MRI scan and calculation of the lesion volume. Number of participants with change in white matter and demyelination on Day 10 compared to Day 1, Day 60 compared to Day 1 and Day 60 compared to Day 10 were reported.
Time Frame: Up to Day 60
Population: All Subjects population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK249320 1 mg/kg | GSK249320 5 mg/kg | GSK249320 15 mg/kg
Number analyzed (Participants) | 17 | 8 | 9 | 8
Participants
  White matter change, Day 10 compared to Day 1 | 9 | 5 | 5 | 2
  White matter change, Day 60 compared to Day 1 | 6 | 6 | 2 | 3
  White matter change, Day 60 compared to Day 10 | 5 | 5 | 1 | 3
  Demyelination, Day 10 compared to Day 1, Yes | 1 | 0 | 3 | 0
  Demyelination, Day 10 compared to Day 1, No | 13 | 8 | 6 | 7
  Demyelination, Day 60 compared to Day 1, No | 14 | 8 | 9 | 6
  Demyelination, Day 60 compared to Day 10, No | 14 | 8 | 9 | 6
  Demyelination, During Study, Yes | 2 | 0 | 3 | 0
  Demyelination, During Study, No | 13 | 8 | 6 | 7

6. Primary Outcome: Number of Participants With Abnormal Clinical Chemistry Parameters
Description: The clinical chemistry parameters analyzed were albumin, calcium, creatinine, glucose, potassium, sodium, total CO2, alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, and total bilirubin. Only those parameters for which at least one abnormal value was reported are summarized. The number of participants with abnormal clinical chemistry findings at specified visit were reported.
Time Frame: Up to Day 112
Population: All Subjects population. Data for only those participants available at the indicated time points were collected and analyzed. Data points with null value for participants analyzed indicate data not collected for respective category and treatment arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK249320 1 mg/kg | GSK249320 5 mg/kg | GSK249320 15 mg/kg
Number analyzed (Participants) | 17 | 8 | 9 | 8
Participants
  Albumin, Visit1 , Day 1, Pre-dose, Low: number analyzed (Participants) | 16 | 8 | 9 | 8
  Albumin, Visit1 , Day 1, Pre-dose, Low | 1 | 0 | 0 | 1
  Albumin, Visit 2 , Day 5, Low: number analyzed (Participants) | 14 | 7 | 9 | 8
  Albumin, Visit 2 , Day 5, Low | 0 | 0 | 0 | 1
  Albumin, Visit 3 , Day 10, Pre-dose, Low: number analyzed (Participants) | 13 | 8 | 8 | 7
  Albumin, Visit 3 , Day 10, Pre-dose, Low | 0 | 0 | 0 | 1
  Albumin, Visit 3 , Day 10, 3 hour, Low: number analyzed (Participants) | 14 | 7 | 8 | 7
  Albumin, Visit 3 , Day 10, 3 hour, Low | 0 | 0 | 0 | 1
  Albumin, Visit 5 , Day 60, Low: number analyzed (Participants) | 14 | 8 | 9 | 6
  Albumin, Visit 5 , Day 60, Low | 0 | 0 | 0 | 1
  ALT, visit 4, day 30, high: number analyzed (Participants) | 13 | 8 | 8 | 6
  ALT, visit 4, day 30, high | 0 | 0 | 1 | 0
  ALT, Visit 6, Day 90, High: number analyzed (Participants) | 14 | 7 | 8 | 6
  ALT, Visit 6, Day 90, High | 0 | 0 | 0 | 1
  ALT, Visit 7, Day 112, High: number analyzed (Participants) | 14 | 8 | 8 | 6
  ALT, Visit 7, Day 112, High | 0 | 0 | 0 | 1
  AST, Visit 4, Day 30, High: number analyzed (Participants) | 13 | 8 | 8 | 6
  AST, Visit 4, Day 30, High | 1 | 0 | 1 | 0
  AST, Visit 6, Day 90, High: number analyzed (Participants) | 14 | 7 | 8 | 5
  AST, Visit 6, Day 90, High | 0 | 0 | 0 | 1
  AST, Visit 7, Day 112, High: number analyzed (Participants) | 14 | 8 | 8 | 5
  AST, Visit 7, Day 112, High | 0 | 0 | 0 | 1
  Calcium, Visit1 , Day 1, Pre-dose, Low: number analyzed (Participants) | 15 | 8 | 9 | 8
  Calcium, Visit1 , Day 1, Pre-dose, Low | 2 | 0 | 1 | 1
  Calcium, Visit1 , Day 1, 24 hour, Low: number analyzed (Participants) | 15 | 7 | 7 | 6
  Calcium, Visit1 , Day 1, 24 hour, Low | 1 | 1 | 1 | 0
  CO2, Visit 1, Day 1, Pre-dose, Low: number analyzed (Participants) | 16 | 8 | 9 | 8
  CO2, Visit 1, Day 1, Pre-dose, Low | 5 | 3 | 6 | 5
  CO2, Visit 1, Day 1, 24 hour, Low: number analyzed (Participants) | 15 | 7 | 7 | 7
  CO2, Visit 1, Day 1, 24 hour, Low | 3 | 3 | 1 | 3
  CO2, Visit 2, Day 5, Low: number analyzed (Participants) | 14 | 7 | 9 | 8
  CO2, Visit 2, Day 5, Low | 3 | 1 | 3 | 4
  CO2, Visit 3, Day 10, Pre-dose, Low: number analyzed (Participants) | 13 | 8 | 8 | 7
  CO2, Visit 3, Day 10, Pre-dose, Low | 2 | 0 | 1 | 2
  CO2, Visit 3, Day 10, 3H, Low: number analyzed (Participants) | 14 | 7 | 8 | 7
  CO2, Visit 3, Day 10, 3H, Low | 3 | 0 | 1 | 1
  CO2, Visit 4, Day 30, Low: number analyzed (Participants) | 13 | 8 | 8 | 6
  CO2, Visit 4, Day 30, Low | 2 | 1 | 2 | 1
  CO2, Visit 5, Day 60, Low: number analyzed (Participants) | 14 | 8 | 9 | 6
  CO2, Visit 5, Day 60, Low | 1 | 0 | 1 | 0
  CO2, Visit 6, Day 90, Low: number analyzed (Participants) | 14 | 7 | 8 | 5
  CO2, Visit 6, Day 90, Low | 2 | 1 | 0 | 0
  CO2, Visit 7, Day 112, Low: number analyzed (Participants) | 14 | 8 | 8 | 6
  CO2, Visit 7, Day 112, Low | 4 | 1 | 0 | 1
  CO2, Early Withdrawal, Low: number analyzed (Participants) | 2 | 0 | 0 | 0
  CO2, Early Withdrawal, Low | 1 |  |  |
  Creatinine, Visit1 , Day 1, Pre-dose, High: number analyzed (Participants) | 15 | 8 | 9 | 8
  Creatinine, Visit1 , Day 1, Pre-dose, High | 0 | 0 | 1 | 0
  Creatinine, Visit 2 , Day 5, High: number analyzed (Participants) | 14 | 7 | 9 | 8
  Creatinine, Visit 2 , Day 5, High | 0 | 0 | 1 | 0
  Creatinine, Visit 3, Day 10, Pre-dose, High: number analyzed (Participants) | 13 | 8 | 8 | 7
  Creatinine, Visit 3, Day 10, Pre-dose, High | 0 | 0 | 1 | 1
  Creatinine, Visit 3, Day 10, 3 hour, High: number analyzed (Participants) | 13 | 7 | 8 | 7
  Creatinine, Visit 3, Day 10, 3 hour, High | 0 | 0 | 1 | 1
  Creatinine, Visit 4, Day 30, High: number analyzed (Participants) | 13 | 8 | 8 | 6
  Creatinine, Visit 4, Day 30, High | 0 | 0 | 1 | 0
  Creatinine, Visit 5, Day 60, High: number analyzed (Participants) | 14 | 8 | 8 | 6
  Creatinine, Visit 5, Day 60, High | 0 | 0 | 1 | 0
  Creatinine, Visit 6 Day 90, High: number analyzed (Participants) | 14 | 7 | 8 | 6
  Creatinine, Visit 6 Day 90, High | 0 | 0 | 1 | 0
  Glucose, Visit 1, Day 1, Pre-dose, High: number analyzed (Participants) | 16 | 8 | 9 | 8
  Glucose, Visit 1, Day 1, Pre-dose, High | 0 | 0 | 2 | 1
  Glucose, Visit 1, Day 1, Pre-dose, Low: number analyzed (Participants) | 16 | 8 | 9 | 8
  Glucose, Visit 1, Day 1, Pre-dose, Low | 0 | 0 | 1 | 0
  Glucose, Visit 1, Day 1, 24 hour, High: number analyzed (Participants) | 15 | 7 | 7 | 7
  Glucose, Visit 1, Day 1, 24 hour, High | 3 | 0 | 1 | 3
  Glucose, Visit 1, Day 1, 24 hour, Low: number analyzed (Participants) | 15 | 7 | 7 | 7
  Glucose, Visit 1, Day 1, 24 hour, Low | 1 | 0 | 0 | 0
  Glucose, Visit 2, Day 5, High: number analyzed (Participants) | 14 | 7 | 9 | 8
  Glucose, Visit 2, Day 5, High | 2 | 0 | 2 | 1
  Glucose, Visit 3, Day 10, Pre-dose, High: number analyzed (Participants) | 13 | 8 | 8 | 6
  Glucose, Visit 3, Day 10, Pre-dose, High | 2 | 0 | 2 | 0
  Glucose, Visit 3, Day 10, 3 hour, High: number analyzed (Participants) | 13 | 7 | 8 | 7
  Glucose, Visit 3, Day 10, 3 hour, High | 1 | 0 | 1 | 1
  Glucose, Visit 4, Day 30, High: number analyzed (Participants) | 13 | 8 | 8 | 6
  Glucose, Visit 4, Day 30, High | 0 | 0 | 1 | 1
  Glucose, Visit 5, Day 60, High: number analyzed (Participants) | 14 | 8 | 9 | 6
  Glucose, Visit 5, Day 60, High | 0 | 1 | 2 | 0
  Glucose, Visit 6, Day 90, High: number analyzed (Participants) | 14 | 7 | 8 | 6
  Glucose, Visit 6, Day 90, High | 0 | 1 | 0 | 0
  Glucose, Visit 7, Day 112, High: number analyzed (Participants) | 14 | 8 | 8 | 6
  Glucose, Visit 7, Day 112, High | 0 | 1 | 1 | 0
  Potassium, Visit 1, Day 1, 24 hour, High: number analyzed (Participants) | 15 | 7 | 7 | 7
  Potassium, Visit 1, Day 1, 24 hour, High | 2 | 0 | 0 | 0
  Potassium, Visit 3, Day 10, Pre-dose, High: number analyzed (Participants) | 13 | 8 | 8 | 7
  Potassium, Visit 3, Day 10, Pre-dose, High | 1 | 0 | 0 | 1
  Potassium, Visit 5, Day 60, High: number analyzed (Participants) | 14 | 8 | 9 | 6
  Potassium, Visit 5, Day 60, High | 0 | 0 | 1 | 0
  Sodium, Visit 2, Day 5, Low: number analyzed (Participants) | 14 | 7 | 9 | 8
  Sodium, Visit 2, Day 5, Low | 1 | 0 | 0 | 0
  Sodium, Visit 3, Day 10, 3 hour, Low: number analyzed (Participants) | 14 | 7 | 8 | 7
  Sodium, Visit 3, Day 10, 3 hour, Low | 1 | 0 | 0 | 0
  Sodium, Visit 4, Day 30, Low: number analyzed (Participants) | 13 | 8 | 8 | 6
  Sodium, Visit 4, Day 30, Low | 1 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Abnormal Hematological Parameters
Description: The clinical chemistry parameters analyzed were white blood cell count, neutrophil count, hemoglobin, platelet count, lymphocytes. Only those parameters for which at least one abnormal value was reported are summarized. The number of participants with abnormal hematology findings at specified visit were reported.
Time Frame: Up to Day 112
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK249320 1 mg/kg | GSK249320 5 mg/kg | GSK249320 15 mg/kg
Number analyzed (Participants) | 17 | 8 | 9 | 8
Participants
  Lymphocytes, Visit 1, Day 1, Pre-dose, Low: number analyzed (Participants) | 16 | 8 | 8 | 8
  Lymphocytes, Visit 1, Day 1, Pre-dose, Low | 0 | 0 | 1 | 0
  Lymphocytes, Visit 1, Day 1, 24 hour, Low: number analyzed (Participants) | 14 | 7 | 9 | 7
  Lymphocytes, Visit 1, Day 1, 24 hour, Low | 0 | 0 | 1 | 0
  Lymphocytes, Visit 2, Day 5, Low: number analyzed (Participants) | 13 | 7 | 9 | 8
  Lymphocytes, Visit 2, Day 5, Low | 1 | 0 | 0 | 0
  Lymphocytes, Visit 6, Day 90, Low: number analyzed (Participants) | 13 | 8 | 8 | 6
  Lymphocytes, Visit 6, Day 90, Low | 1 | 0 | 0 | 0
  Lymphocytes, Visit 7, Day 112, Low: number analyzed (Participants) | 13 | 8 | 7 | 6
  Lymphocytes, Visit 7, Day 112, Low | 1 | 0 | 0 | 0
  Lymphocytes, Early withdrawal, Low: number analyzed (Participants) | 2 | 0 | 0 | 0
  Lymphocytes, Early withdrawal, Low | 1 |  |  |
  Total Neutrophils, Visit 5, Day 60, Low: number analyzed (Participants) | 14 | 8 | 9 | 6
  Total Neutrophils, Visit 5, Day 60, Low | 1 | 0 | 0 | 0
  Total Neutrophils, Visit 6, Day 90, Low: number analyzed (Participants) | 13 | 8 | 8 | 6
  Total Neutrophils, Visit 6, Day 90, Low | 1 | 0 | 0 | 0
  Platelet count, Visit 4, Day 30, High: number analyzed (Participants) | 13 | 8 | 8 | 7
  Platelet count, Visit 4, Day 30, High | 1 | 0 | 0 | 0
  Platelet count, Visit 5, Day 60, High: number analyzed (Participants) | 13 | 8 | 8 | 7
  Platelet count, Visit 5, Day 60, High | 1 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Positive Antibodies to GSK249320
Description: Presence of antibodies to GSK249320 were assessed in serum samples of participants using immunoelectro-chemiluminescent assay. Number of participants with positive antibodies to GSK249320 were reported. Only visits where the true positive antibody detection was observed were reported.
Time Frame: Day 1, 5, 10, 30, 60, 90 and 112
Population: All Subjects population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK249320 1 mg/kg | GSK249320 5 mg/kg | GSK249320 15 mg/kg
Number analyzed (Participants) | 17 | 8 | 9 | 8
Participants
  Visit 1 Day 1 True positive | 0 | 0 | 1 | 0
  Visit 3 Day 10 True positive: number analyzed (Participants) | 13 | 8 | 9 | 7
  Visit 3 Day 10 True positive | 0 | 1 | 1 | 0
  Visit 4 Day 30 True positive: number analyzed (Participants) | 14 | 8 | 9 | 7
  Visit 4 Day 30 True positive | 0 | 0 | 1 | 0
  Visit 5 Day 60 True positive: number analyzed (Participants) | 14 | 8 | 8 | 7
  Visit 5 Day 60 True positive | 0 | 0 | 1 | 0

9. Secondary Outcome: Mean Area Under the Concentration-time Curve From Time Zero (Pre-dose) Extrapolated to Infinite Time (AUC 0-inf) and Area Under the Concentration-time Curve From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration (AUC0-t)
Description: The pharmacokinetic parameters were calculated by standard non-compartmental analysis using Win Nonlin Pro 4.1. All calculations of non-compartmental parameters were based on actual sampling times. AUC0-t was determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations. AUC(0-inf) were calculated, where data permit, as the sum of area under the concentration-time curve over the dosing interval from 0 to Day 10 ±1 day (AUC0-10d) and C10d/z, where C10d is the observed plasma concentration at day 10 and z is the terminal phase rate constant calculated after the second dose.
Time Frame: Day 1 (Pre-dose, 1, 3, 6, 12 and 24 hour) and Day 10 (Pre-dose, 1, 3 hour)
Population: Pharmacokinetic population comprised of participants from the 'All Subjects' population for whom a pharmacokinetic sample was obtained and analyzed. Only those participants with data available for analysis were analyzed.
Measure: Mean (Standard Deviation); unit: Hour*mg/millilitre (mL)
Arm/Group | GSK249320 1 mg/kg | GSK249320 5 mg/kg | GSK249320 15 mg/kg
Number analyzed (Participants) | 8 | 9 | 8
Hour*mg/millilitre (mL)
  AUC(0-inf): number analyzed (Participants) | 8 | 8 | 7
  AUC(0-inf) | 15.20 (4.049) | 71.01 (14.426) | 192.88 (75.413)
  AUC(0-t), Dose 1: number analyzed (Participants) | 8 | 8 | 8
  AUC(0-t), Dose 1 | 4.12 (0.643) | 17.25 (3.704) | 51.07 (18.719)
  AUC(0-t), Dose 2: number analyzed (Participants) | 8 | 8 | 7
  AUC(0-t), Dose 2 | 25.64 (7.272) | 118.38 (28.885) | 365.63 (83.891)

10. Secondary Outcome: Mean Maximum Observed Concentration (Cmax) and Last Observed Quantifiable Concentration (Ct)
Description: The pharmacokinetic parameters were calculated by standard non- compartmental analysis using Win Nonlin Pro 4.1. All calculations of non-compartmental parameters were based on actual sampling times. Cmax and Ct were determined directly from the raw concentration-time data.
Time Frame: Day 1 (Pre-dose, 1, 3, 6, 12 and 24 hour) and Day 10 (Pre-dose, 1, 3 hour)
Population: Pharmacokinetic population. Only those participants with data available for analysis were analyzed.
Measure: Mean (Standard Deviation); unit: microgram (ug) per mL
Arm/Group | GSK249320 1 mg/kg | GSK249320 5 mg/kg | GSK249320 15 mg/kg
Number analyzed (Participants) | 8 | 9 | 8
microgram (ug) per mL
  Cmax, Dose 1: number analyzed (Participants) | 8 | 8 | 8
  Cmax, Dose 1 | 38.62 (8.832) | 157.42 (25.814) | 508.20 (74.468)
  Cmax, Dose 2: number analyzed (Participants) | 8 | 8 | 7
  Cmax, Dose 2 | 53.06 (17.650) | 215.71 (30.617) | 756.98 (178.150)
  Ct, Dose 1 | 14.9528 (3.63064) | 59.3422 (22.10706) | 192.1709 (92.75262)
  Ct, Dose 2: number analyzed (Participants) | 8 | 9 | 7
  Ct, Dose 2 | 0.6647 (0.35900) | 6.8148 (4.04066) | 22.1555 (17.84140)

11. Secondary Outcome: Mean Time of Occurrence of Cmax (Tmax) and Time of Last Observed Quantifiable Concentration (Tlast)
Description: The pharmacokinetic parameters were calculated by standard non-compartmental analysis using Win Nonlin Pro 4.1. All calculations of non-compartmental parameters were based on actual sampling times. Tmax and tlast were determined directly from the raw concentration-time data.
Time Frame: Day 1 (Pre-dose, 1, 3, 6, 12 and 24 hour) and Day 10 (Pre-dose, 1, 3 hour)
Population: Pharmacokinetics population. Only those participants with data available for analysis were analyzed.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | GSK249320 1 mg/kg | GSK249320 5 mg/kg | GSK249320 15 mg/kg
Number analyzed (Participants) | 8 | 9 | 8
hour
  tmax, Dose 1 | 2.723 (3.8135) | 1.807 (1.7017) | 1.885 (1.8745)
  tmax, Dose 2: number analyzed (Participants) | 8 | 9 | 7
  tmax, Dose 2 | 2.013 (1.0562) | 1.618 (1.1276) | 1.874 (1.0792)
  tlast, Dose 1 | 207.43 (26.247) | 192.67 (39.911) | 205.47 (83.950)
  tlast, Dose 2: number analyzed (Participants) | 8 | 9 | 7
  tlast, Dose 2 | 2901.11 (144.034) | 2539.06 (418.783) | 2403.84 (141.350)

12. Secondary Outcome: Mean Terminal Phase Half-life (t1/2)
Description: The pharmacokinetic parameters were calculated by standard non-compartmental analysis using Win Nonlin Pro 4.1. All calculations of non-compartmental parameters were based on actual sampling times. The apparent t1/2 obtained as the ratio of natural log (ln)^2/ lambda-Z, where lambda-Z is the terminal phase rate constant estimated by linear regression analysis of the log transformed concentration-time data.
Time Frame: Day 1 (Pre-dose, 1, 3, 6, 12 and 24 hour) and Day 10 (Pre-dose, 1, 3 hour)
Population: Pharmacokinetics population. Only those participants with data available for analysis were analyzed.
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | GSK249320 1 mg/kg | GSK249320 5 mg/kg | GSK249320 15 mg/kg
Number analyzed (Participants) | 8 | 9 | 8
Day | 21.11 (3.121) | 24.01 (5.240) | 24.01 (8.551)

13. Secondary Outcome: Mean Terminal Phase Rate Constant ( Lambda-Z)
Description: The pharmacokinetic parameters were calculated by standard non-compartmental analysis using Win Nonlin Pro 4.1. All calculations of non-compartmental parameters were based on actual sampling times. Lambda-Z is the terminal phase rate constant estimated by linear regression analysis of the log transformed concentration-time data.
Time Frame: Day 1 (Pre-dose, 1, 3, 6, 12 and 24 hour) and Day 10 (Pre-dose, 1, 3 hour)
Population: Pharmacokinetics population. Only those participants with data available for analysis were analyzed.
Measure: Mean (Standard Deviation); unit: 1/ hour
Arm/Group | GSK249320 1 mg/kg | GSK249320 5 mg/kg | GSK249320 15 mg/kg
Number analyzed (Participants) | 8 | 9 | 8
1/ hour
  lambda-z, Dose 1: number analyzed (Participants) | 8 | 9 | 7
  lambda-z, Dose 1 | 0.00138 (0.000191) | 0.00126 (0.000292) | 0.00130 (0.000327)
  lambda-z, Dose 2: number analyzed (Participants) | 8 | 9 | 7
  lambda-z, Dose 2 | 0.00139 (0.000207) | 0.00126 (0.000281) | 0.00130 (0.000327)

14. Secondary Outcome: Mean Clearance of GSK249320
Description: The pharmacokinetic parameters were calculated by standard non-compartmental analysis using Win Nonlin Pro 4.1. All calculations of non-compartmental parameters were based on actual sampling times. The clearance was calculated as Dose/ AUC(0-inf).
Time Frame: Day 1 (Pre-dose, 1, 3, 6, 12 and 24 hour) and Day 10 (Pre-dose, 1, 3 hour)
Population: Pharmacokinetics population. Only those participants with data available for analysis were analyzed.
Measure: Mean (Standard Deviation); unit: mL/hour/killogram (kg)
Arm/Group | GSK249320 1 mg/kg | GSK249320 5 mg/kg | GSK249320 15 mg/kg
Number analyzed (Participants) | 8 | 9 | 7
mL/hour/killogram (kg) | 0.0700 (0.01835) | 0.0750 (0.01545) | 0.0886 (0.03652)

15. Secondary Outcome: Mean Change in Mean Gait Velocity
Description: Gait velocity is an objective, quantitative, reliable, valid and sensitive measure of lower extremity motor recovery in the stroke population. Changes in gait velocity correlates with physical functioning and quality of life. Gait velocity was assessed over a level, indoor 10 meter distance. The time (in seconds) it takes the participant to travel the 10 meter distance was recorded. Participants was asked to walk at their usual or normal pace and may use their normal assistive devices. Baseline assessments were recorded at Day 5 of the study. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. If either the Baseline or post-randomization value was missing, the change from Baseline was set to missing as well.
Time Frame: Baseline (Day 5), Day 30, 60, 90, 112
Population: All Subjects population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Meters/second
Arm/Group | Placebo | GSK249320 1 mg/kg | GSK249320 5 mg/kg | GSK249320 15 mg/kg
Number analyzed (Participants) | 17 | 8 | 9 | 8
Meters/second
  Visit 4 Day 30: number analyzed (Participants) | 13 | 7 | 9 | 6
  Visit 4 Day 30 | -0.010 (0.4021) | 0.548 (0.6015) | 0.649 (0.6114) | 0.210 (0.3957)
  Visit 5 Day 60: number analyzed (Participants) | 12 | 8 | 9 | 6
  Visit 5 Day 60 | 0.252 (0.4005) | 0.679 (0.7587) | 0.730 (0.8277) | 0.203 (0.7378)
  Visit 6 Day 90: number analyzed (Participants) | 13 | 8 | 8 | 5
  Visit 6 Day 90 | 0.207 (0.3327) | 0.925 (0.7199) | 0.539 (0.7267) | 0.302 (0.4770)
  Visit 7 Day 112: number analyzed (Participants) | 12 | 8 | 7 | 5
  Visit 7 Day 112 | 0.376 (0.4164) | 1.052 (0.6678) | 1.047 (0.8208) | 0.408 (0.5011)
Statistical Analysis 1: Comparison: Placebo vs GSK249320 1 mg/kg; Placebo Vs GSK249320 1 mg/kg, Visit 4; Test type: Superiority or Other; Mixed Model Repeated Measure Analysis; Mean Difference (Net) = 0.45, 95% CI 2-sided [-0.03 to 0.92], Standard Error of Mean 0.231 — Mean difference = GSK249320 1 mg/kg - Placebo
Statistical Analysis 2: Comparison: Placebo vs GSK249320 5 mg/kg; Placebo Vs GSK249320 5 mg/kg, Visit 4; Test type: Superiority or Other; Mixed Model Repeated Measure Analysis; Mean Difference (Net) = 0.69, 95% CI 2-sided [0.25 to 1.13], Standard Error of Mean 0.214 — Mean difference = GSK249320 5 mg/kg - Placebo
Statistical Analysis 3: Comparison: Placebo vs GSK249320 15 mg/kg; Placebo Vs GSK249320 15 mg/kg, Visit 4; Test type: Superiority or Other; Mixed Model Repeated Measure Analysis; Mean Difference (Net) = 0.30, 95% CI 2-sided [-0.20 to 0.80], Standard Error of Mean 0.246 — Mean difference= GSK249320 15 mg/kg - Placebo
Statistical Analysis 4: Comparison: Placebo vs GSK249320 1 mg/kg; Placebo Vs GSK249320 1 mg/kg, Visit 5; Test type: Superiority or Other; Mixed Model Repeated Measure Analysis; Mean Difference (Net) = 0.35, 95% CI 2-sided [-0.24 to 0.95], Standard Error of Mean 0.292 — Mean difference= GSK249320 1 mg/kg - Placebo
Statistical Analysis 5: Comparison: Placebo vs GSK249320 5 mg/kg; Placebo Vs GSK249320 5 mg/kg, Visit 5; Test type: Superiority or Other; Mixed Model Repeated Measure Analysis; Mean Difference (Net) = 0.52, 95% CI 2-sided [-0.05 to 1.09], Standard Error of Mean 0.279 — Mean difference= GSK249320 5 mg/kg- Placebo
Statistical Analysis 6: Comparison: Placebo vs GSK249320 15 mg/kg; Placebo Vs GSK249320 15 mg/kg, Visit 5; Test type: Superiority or Other; Mixed Model Repeated Measure Analysis; Mean Difference (Net) = 0.04, 95% CI 2-sided [-0.61 to 0.69], Standard Error of Mean 0.319 — Mean difference= GSK249320 15 mg/kg - Placebo
Statistical Analysis 7: Comparison: Placebo vs GSK249320 1 mg/kg; Placebo Vs GSK249320 1 mg/kg, Visit 6; Test type: Superiority or Other; Mixed Model Repeated Measure Analysis; Mean Difference (Net) = 0.63, 95% CI 2-sided [0.15 to 1.11], Standard Error of Mean 0.235 — Mean difference= GSK249320 1 mg/kg - Placebo
Statistical Analysis 8: Comparison: Placebo vs GSK249320 5 mg/kg; Placebo Vs GSK249320 5 mg/kg, Visit 6; Test type: Superiority or Other; Mixed Model Repeated Measure Analysis; Mean Difference (Net) = 0.40, 95% CI 2-sided [-0.06 to 0.86], Standard Error of Mean 0.225 — Mean difference= GSK249320 5 mg/kg - Placebo
Statistical Analysis 9: Comparison: Placebo vs GSK249320 15 mg/kg; Placebo Vs GSK249320 15 mg/kg, Visit 6; Test type: Superiority or Other; Mixed Model Repeated Measure Analysis; Mean Difference (Net) = 0.24, 95% CI 2-sided [-0.29 to 0.77], Standard Error of Mean 0.259 — Mean difference= GSK249320 15 mg/kg - Placebo
Statistical Analysis 10: Comparison: Placebo vs GSK249320 1 mg/kg; Placebo Vs GSK249320 1 mg/kg, Visit 7; Test type: Superiority or Other; Mixed Model Repeated Measure Analysis; Mean Difference (Net) = 0.61, 95% CI 2-sided [0.10 to 1.12], Standard Error of Mean 0.251 — Mean difference= GSK249320 1 mg/kg - Placebo
Statistical Analysis 11: Comparison: Placebo vs GSK249320 5 mg/kg; Placebo Vs GSK249320 5 mg/kg, Visit 7; Test type: Superiority or Other; Mixed Model Repeated Measure Analysis; Mean Difference (Net) = 0.59, 95% CI 2-sided [0.09 to 1.08], Standard Error of Mean 0.242 — Mean difference= GSK249320 5 mg/kg - Placebo
Statistical Analysis 12: Comparison: Placebo vs GSK249320 15 mg/kg; Placebo Vs GSK249320 5 mg/kg, Visit 7; Test type: Superiority or Other; Mixed Model Repeated Measure Analysis; Mean Difference (Net) = 0.17, 95% CI 2-sided [-0.39 to 0.73], Standard Error of Mean 0.277 — Mean difference= GSK249320 15 mg/kg - Placebo

16. Secondary Outcome: Mean Change in Berg Balance Scale (BBS) Total Score
Description: BBS is a performance based measure of balance. It is reliable, valid and responsive to change in the stroke population. BBS is a staff-assessed measure that requires the participant to perform 14 activities that evaluate ability to maintain balance. The BBS typically takes 10-15minute to complete. Participants were not allowed to use assistive devices while performing the activities. Each activity was evaluated by direct observation of the participant's performance and was scored on a 5-point ordinal scale (0-4) where a score of 0 represents inability to perform the activity and a score of 4 represents independence in the activity. The minimum total score on the BBS was 0 and maximum was 56. Baseline assessments were recorded at Day 5 of the study. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. If either the Baseline or post-randomization value was missing, the change from Baseline was set to missing as well.
Time Frame: Baseline (Day 5), Day 30, 60, 90 and 112
Population: All Subjects population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on Scale
Arm/Group | Placebo | GSK249320 1 mg/kg | GSK249320 5 mg/kg | GSK249320 15 mg/kg
Number analyzed (Participants) | 17 | 8 | 9 | 8
Score on Scale
  Visit 4 Day 30: number analyzed (Participants) | 13 | 8 | 9 | 6
  Visit 4 Day 30 | 6.8 (14.35) | 17.5 (12.94) | 14.8 (17.05) | 5.7 (10.25)
  Visit 5 Day 60: number analyzed (Participants) | 13 | 7 | 9 | 5
  Visit 5 Day 60 | 10.7 (16.29) | 21.7 (18.83) | 19.0 (17.78) | 12.2 (18.58)
  Visit 6 Day 90: number analyzed (Participants) | 13 | 8 | 8 | 5
  Visit 6 Day 90 | 13.5 (16.47) | 24.4 (18.88) | 20.4 (19.94) | -0.2 (6.72)
  Visit 7 Day 112: number analyzed (Participants) | 13 | 8 | 7 | 5
  Visit 7 Day 112 | 14.6 (18.75) | 25.4 (20.56) | 24.7 (18.96) | 11.8 (18.12)
Statistical Analysis 1: Comparison: Placebo vs GSK249320 1 mg/kg; Placebo Vs GSK249320 1 mg/kg, visit 4; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 9.56, 95% CI 2-sided [-0.60 to 19.71], Standard Error of Mean 4.981 — Mean difference =GSK249320 1 mg/kg - Placebo
Statistical Analysis 2: Comparison: Placebo vs GSK249320 5 mg/kg; Placebo Vs GSK249320 5 mg/kg, Visit 4; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 8.47, 95% CI 2-sided [-1.32 to 18.26], Standard Error of Mean 4.801 — Mean difference= GSK249320 5 mg/kg - Placebo
Statistical Analysis 3: Comparison: Placebo vs GSK249320 15 mg/kg; Placebo Vs GSK249320 15 mg/kg, Visit 4; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Median Difference (Final Values) = 0.09, 95% CI 2-sided [-11.1 to 11.24], Standard Error of Mean 5.470 — Mean difference= GSK249320 GSK249320 15 mg/kg - Placebo
Statistical Analysis 4: Comparison: Placebo vs GSK249320 1 mg/kg; Placebo Vs GSK249320 1 mg/kg, Visit 5; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 11.58, 95% CI 2-sided [0.01 to 23.15], Standard Error of Mean 5.631 — Mean difference= GSK249320 1 mg/kg - Placebo
Statistical Analysis 5: Comparison: Placebo vs GSK249320 5 mg/kg; Placebo Vs GSK249320 5 mg/kg, Visit 5; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 8.77, 95% CI 2-sided [-2.35 to 19.89], Standard Error of Mean 5.411 — Mean difference= GSK249320 5 mg/kg - Placebo
Statistical Analysis 6: Comparison: Placebo vs GSK249320 15 mg/kg; Placebo Vs GSK249320 15 mg/kg, Visit 5; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Final Values) = 0.49, 95% CI 2-sided [-12.2 to 13.21], Standard Error of Mean 6.195 — Mean difference= GSK249320 15 mg/kg - Placebo
Statistical Analysis 7: Comparison: Placebo vs GSK249320 1 mg/kg; Placebo Vs GSK249320 1 mg/kg, Visit 6; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 9.66, 95% CI 2-sided [-1.34 to 20.66], Standard Error of Mean 5.351 — Mean difference= GSK249320 1 mg/kg - Placebo
Statistical Analysis 8: Comparison: Placebo vs GSK249320 5 mg/kg; Placebo Vs GSK249320 5 mg/kg, Visit 6; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 7.45, 95% CI 2-sided [-3.22 to 18.13], Standard Error of Mean 5.198 — Mean difference= GSK249320 5 mg/kg - Placebo
Statistical Analysis 9: Comparison: Placebo vs GSK249320 15 mg/kg; Placebo Vs GSK249320 15 mg/kg, Visit 6; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = -10.63, 95% CI 2-sided [-22.9 to 1.60], Standard Error of Mean 5.959 — Mean difference= GSK249320 15 mg/kg - Placebo
Statistical Analysis 10: Comparison: Placebo vs GSK249320 1 mg/kg; Placebo Vs GSK249320 1 mg/kg, visit 7; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 9.59, 95% CI 2-sided [-3.07 to 22.24], Standard Error of Mean 6.134 — Mean difference= GSK249320 1 mg/kg - Placebo
Statistical Analysis 11: Comparison: Placebo vs GSK249320 5 mg/kg; Placebo Vs GSK249320 5 mg/kg, Visit 7; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 5.89, 95% CI 2-sided [-6.37 to 18.15], Standard Error of Mean 5.948 — Mean difference= GSK249320 5 mg/kg - Placebo
Statistical Analysis 12: Comparison: Placebo vs GSK249320 15 mg/kg; Placebo Vs GSK249320 15 mg/kg, Visit 7; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = -3.11, 95% CI 2-sided [-17.1 to 10.84], Standard Error of Mean 6.768 — Mean difference= GSK249320 15 mg/kg - Placebo

17. Secondary Outcome: Mean Change in Total Fugl-Meyer Motor (FM) Assessment
Description: The FM assessment is a staff-assessed, disease specific, quantitative measure of impairment that is used to assess recovery of sensorimotor function post stroke. The FM is designed to assess the domains of motor function, balance, sensation and joint function. For this study, only the motor function domain was assessed. The motor domain scale takes approximately 30 minutes to complete and evaluates both the upper and lower extremities by direct observation of the participant's performance of 50 items that measure movement, coordination, and reflex action. Each item was scored from 0-2 for a minimum total score of 0 (hemiplegia) and a maximum total score of 100 (normal motor performance). Baseline assessments were recorded at Day 5 of the study. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. If either the Baseline or post-randomization value was missing, the change from Baseline was set to missing as well.
Time Frame: Baseline (Day 5), Day 30 and 112
Population: All subjects population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on Scale
Arm/Group | Placebo | GSK249320 1 mg/kg | GSK249320 5 mg/kg | GSK249320 15 mg/kg
Number analyzed (Participants) | 17 | 8 | 9 | 8
Score on Scale
  Total Score, Visit 4 Day 30: number analyzed (Participants) | 14 | 8 | 9 | 7
  Total Score, Visit 4 Day 30 | 10.2 (19.19) | 8.8 (10.51) | 17.0 (18.23) | 3.1 (21.56)
  Total Score, Visit 7 Day 112: number analyzed (Participants) | 14 | 8 | 7 | 6
  Total Score, Visit 7 Day 112 | 19.6 (23.13) | 17.3 (20.96) | 25.3 (28.40) | 8.7 (34.59)
Statistical Analysis 1: Comparison: Placebo vs GSK249320 1 mg/kg; Placebo Vs GSK249320 1 mg/kg, Visit 4; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = -1.47, 95% CI 2-sided [-15.81 to 12.86], Standard Error of Mean 7.047 — Mean difference= GSK249320 1 mg/kg - Placebo. Change in Total Fugl-Meyer assessment= Treatment + Visit + Treatment * Visit + Baseline
Statistical Analysis 2: Comparison: Placebo vs GSK249320 5 mg/kg; Placebo Vs GSK249320 5 mg/kg, Visit 4; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Median Difference (Net) = 9.86, 95% CI 2-sided [-4.08 to 23.80], Standard Error of Mean 6.852 — Mean difference= GSK249320 5 mg/kg - Placebo. Change in Total Fugl-Meyer assessment= Treatment + Visit + Treatment * Visit + Baseline
Statistical Analysis 3: Comparison: Placebo vs GSK249320 15 mg/kg; Placebo Vs GSK249320 15 mg/kg, Visit 4; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Median Difference (Net) = -5.40, 95% CI 2-sided [-20.41 to 9.60], Standard Error of Mean 7.376 — Mean difference= GSK249320 15 mg/kg - Placebo. Change in Total Fugl-Meyer assessment= Treatment + Visit + Treatment * Visit + Baseline
Statistical Analysis 4: Comparison: Placebo vs GSK249320 1 mg/kg; Placebo Vs GSK249320 1 mg/kg, Visit 7; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Median Difference (Net) = -2.40, 95% CI 2-sided [-22.87 to 18.07], Standard Error of Mean 10.040 — [estimate comment as in outcome 17, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs GSK249320 5 mg/kg; Placebo Vs GSK249320 5 mg/kg, Visit 7; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 5.03, 95% CI 2-sided [-15.95 to 26.00], Standard Error of Mean 10.310 — [estimate comment as in outcome 17, analysis 2]
Statistical Analysis 6: Comparison: Placebo vs GSK249320 15 mg/kg; Placebo Vs GSK249320 15 mg/kg, Visit 7; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Median Difference (Net) = -10.07, 95% CI 2-sided [-32.29 to 12.15], Standard Error of Mean 10.916 — Mean difference= GSK249320 15 mg/kg - Placebo Change in Total Fugl-Meyer assessment= Treatment + Visit + Treatment * Visit + Baseline

18. Secondary Outcome: Mean Change in Total Box and Blocks Transferred on Affected Side
Description: The Box and Blocks test is an objective, gross manual dexterity test that is reliable and valid in individuals with upper limb impairments. Box and Blocks was a staff-assessed, participant completed test that required the participant to move small wooden blocks from one side of a partitioned box to the other. The score was determined by the number of blocks transferred within a 60 second time period. More number of blocks transferred as compared to Baseline indicated improvement. Both the impaired and normal limbs were tested, starting with the normal limb. The number of blocks transferred were recorded. Baseline assessments were recorded at Day 1 of the study. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. If either the Baseline or post-randomization value was missing, the change from Baseline was set to missing as well.
Time Frame: Baseline (Day 1), Day 30, 60, 90 and 112
Population: All subjects population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Blocks
Arm/Group | Placebo | GSK249320 1 mg/kg | GSK249320 5 mg/kg | GSK249320 15 mg/kg
Number analyzed (Participants) | 17 | 8 | 9 | 8
Blocks
  Visit 4 Day 30: number analyzed (Participants) | 14 | 8 | 9 | 7
  Visit 4 Day 30 | 8.5 (11.02) | 8.6 (9.01) | 11.3 (11.30) | 13.0 (13.83)
  Visit 5 Day 60: number analyzed (Participants) | 14 | 8 | 9 | 7
  Visit 5 Day 60 | 13.83 (12.33) | 14.6 (18.45) | 15.6 (13.41) | 10.9 (13.57)
  Visit 6 Day 90: number analyzed (Participants) | 14 | 8 | 8 | 6
  Visit 6 Day 90 | 15.5 (14.11) | 16.1 (15.68) | 18.0 (15.18) | 14.8 (16.50)
  Visit 7 Day 112: number analyzed (Participants) | 14 | 8 | 7 | 6
  Visit 7 Day 112 | 16.5 (14.18) | 18.8 (15.22) | 18.3 (19.67) | 15.2 (15.55)
Statistical Analysis 1: Comparison: Placebo vs GSK249320 1 mg/kg; Placebo Vs GSK249320 1 mg/kg, Visit 4; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 0.13, 95% CI 2-sided [-10.4 to 10.61], Standard Error of Mean 5.147 — Mean difference= GSK249320 1 mg/kg - Placebo Affected Change from Baseline = Treatment + Visit + Treatment * Visit + Affected Baseline + Unaffected Baseline
Statistical Analysis 2: Comparison: Placebo vs GSK249320 5 mg/kg; Placebo Vs GSK249320 5 mg/kg, Visit 4; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 2.75, 95% CI 2-sided [-7.75 to 13.26], Standard Error of Mean 5.157 — Mean difference= GSK249320 5 mg/kg - Placebo Affected Change from Baseline = Treatment + Visit + Treatment * Visit + Affected Baseline + Unaffected Baseline
Statistical Analysis 3: Comparison: Placebo vs GSK249320 15 mg/kg; Placebo Vs GSK249320 15 mg/kg, Visit 4; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 4.85, 95% CI 2-sided [-6.17 to 15.88], Standard Error of Mean 5.409 — Mean difference= GSK249320 15 mg/kg - Placebo Affected Change from Baseline = Treatment + Visit + Treatment * Visit + Affected Baseline + Unaffected Baseline
Statistical Analysis 4: Comparison: Placebo vs GSK249320 1 mg/kg; Placebo Vs GSK249320 1 mg/kg, Visit 5; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 1.20, 95% CI 2-sided [-12.1 to 14.45], Standard Error of Mean 6.504 — [estimate comment as in outcome 18, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs GSK249320 5 mg/kg; Placebo Vs GSK249320 5 mg/kg, Visit 5; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 2.05, 95% CI 2-sided [-11.0 to 15.12], Standard Error of Mean 6.426 — [estimate comment as in outcome 18, analysis 2]
Statistical Analysis 6: Comparison: Placebo vs GSK249320 15 mg/kg; Placebo Vs GSK249320 15 mg/kg, Visit 5; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = -2.22, 95% CI 2-sided [-16.1 to 11.68], Standard Error of Mean 6.820 — [estimate comment as in outcome 18, analysis 3]
Statistical Analysis 7: Comparison: Placebo vs GSK249320 1 mg/kg; Placebo Vs GSK249320 1 mg/kg, Visit 6; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Median Difference (Net) = 0.63, 95% CI 2-sided [-12.9 to 14.18], Standard Error of Mean 6.664 — [estimate comment as in outcome 18, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs GSK249320 5 mg/kg; Placebo Vs GSK249320 5 mg/kg, Visit 6; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 1.03, 95% CI [-12.4 to 14.43], Standard Error of Mean 6.595 — [estimate comment as in outcome 18, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs GSK249320 15 mg/kg; Placebo Vs GSK249320 15 mg/kg, Visit 6; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Median Difference (Net) = -0.95, 95% CI 2-sided [-15.2 to 13.32], Standard Error of Mean 7.020 — [estimate comment as in outcome 18, analysis 3]
Statistical Analysis 10: Comparison: Placebo vs GSK249320 1 mg/kg; Placebo Vs GSK249320 1 mg/kg, Visit 7; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 2.25, 95% CI 2-sided [-11.9 to 16.40], Standard Error of Mean 6.953 — [estimate comment as in outcome 18, analysis 1]
Statistical Analysis 11: Comparison: Placebo vs GSK249320 5 mg/kg; Placebo Vs GSK249320 5 mg/kg, Visit 7; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 3.52, 95% CI 2-sided [-10.5 to 17.55], Standard Error of Mean 6.909 — [estimate comment as in outcome 18, analysis 2]
Statistical Analysis 12: Comparison: Placebo vs GSK249320 15 mg/kg; Placebo Vs GSK249320 15 mg/kg, Visit 7; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = -0.50, 95% CI 2-sided [-15.4 to 14.39], Standard Error of Mean 7.328 — [estimate comment as in outcome 18, analysis 3]

19. Secondary Outcome: Mean Change in Grip Strength on Affected Side
Description: Grip strength is an objective measure of arm motor recovery in stroke participants and correlate with functional status and predict recovery. Grip strength was evaluated by a hand grip dynamometer. Three replicate trials was collected for both the impaired and normal hand, starting with the normal hand. Each trial was separated by a resting period of approximately 15-30 seconds. Participants was instructed to squeeze as hard as possible while using a standardized position of grip and the resulting dynamometer reading (in kg) was recorded. The grip strength measures was conducted within approximately 5 minutes. Baseline assessments were recorded at Day 1 of the study. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. If either the Baseline or post-randomization value was missing, the change from Baseline was set to missing as well.
Time Frame: Baseline (Day 1), Day 30, 60, 90 and 112
Population: All Subjects population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Placebo | GSK249320 1 mg/kg | GSK249320 5 mg/kg | GSK249320 15 mg/kg
Number analyzed (Participants) | 17 | 8 | 9 | 8
Kg
  Visit 4 Day 30: number analyzed (Participants) | 13 | 8 | 8 | 7
  Visit 4 Day 30 | -1.01 (9.291) | 2.94 (5.897) | 1.13 (6.200) | 5.52 (6.526)
  Visit 5 Day 60: number analyzed (Participants) | 14 | 8 | 8 | 7
  Visit 5 Day 60 | 2.64 (11.314) | 5.50 (6.208) | 1.25 (6.791) | 4.57 (7.615)
  Visit 6 Day 90: number analyzed (Participants) | 14 | 8 | 7 | 6
  Visit 6 Day 90 | 2.24 (10.811) | 6.50 (8.118) | 3.71 (8.236) | 4.44 (7.644)
  Visit 7 Day 112: number analyzed (Participants) | 14 | 8 | 6 | 6
  Visit 7 Day 112 | 2.74 (11.824) | 6.58 (7.115) | 1.28 (9.923) | 6.78 (8.334)
Statistical Analysis 1: Comparison: Placebo vs GSK249320 1 mg/kg; Placebo Vs GSK249320 1 mg/kg, Visit 4; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 1.66, 95% CI 2-sided [-5.33 to 8.65], Standard Error of Mean 3.420 — Mean difference= GSK249320 1 mg/kg - Placebo. Affected Change from Baseline = Treatment + Visit + Treatment * Visit + Affected Baseline + Unaffected Baseline
Statistical Analysis 2: Comparison: Placebo vs GSK249320 5 mg/kg; Placebo Vs GSK249320 5 mg/kg, Visit 4; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = -0.30, 95% CI 2-sided [-7.56 to 6.96], Standard Error of Mean 3.550 — Mean difference= GSK249320 5 mg/kg - Placebo. Affected Change from Baseline = Treatment + Visit + Treatment * Visit + Affected Baseline + Unaffected Baseline
Statistical Analysis 3: Comparison: Placebo vs GSK249320 15 mg/kg; Placebo Vs GSK249320 15 mg/kg, Visit 4; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 4.56, 95% CI 2-sided [-2.67 to 11.78], Standard Error of Mean 3.534 — Mean difference= GSK249320 15 mg/kg - Placebo. Affected Change from Baseline = Treatment + Visit + Treatment * Visit + Affected Baseline + Unaffected Baseline
Statistical Analysis 4: Comparison: Placebo vs GSK249320 1 mg/kg; Placebo Vs GSK249320 1 mg/kg, Visit 5; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 2.05, 95% CI 2-sided [-5.78 to 9.89], Standard Error of Mean 3.841 — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs GSK249320 5 mg/kg; Placebo Vs GSK249320 5 mg/kg, Visit 5; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Median Difference (Net) = -2.35, 95% CI 2-sided [-10.4 to 5.72], Standard Error of Mean 3.958 — [estimate comment as in outcome 19, analysis 2]
Statistical Analysis 6: Comparison: Placebo vs GSK249320 15 mg/kg; Placebo Vs GSK249320 15 mg/kg, Visit 5; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 1.44, 95% CI 2-sided [-6.68 to 9.55], Standard Error of Mean 3.978 — [estimate comment as in outcome 19, analysis 3]
Statistical Analysis 7: Comparison: Placebo vs GSK249320 1 mg/kg; Placebo Vs GSK249320 1 mg/kg, Visit 6; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 3.46, 95% CI 2-sided [-4.94 to 11.85], Standard Error of Mean 4.109 — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs GSK249320 5 mg/kg; Placebo Vs GSK249320 5 mg/kg, Visit 6; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 0.49, 95% CI 2-sided [-8.15 to 9.12], Standard Error of Mean 4.235 — [estimate comment as in outcome 19, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs GSK249320 15 mg/kg; Placebo Vs GSK249320 15 mg/kg, Visit 6; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Median Difference (Net) = 0.77, 95% CI 2-sided [-7.97 to 9.50], Standard Error of Mean 4.280 — [estimate comment as in outcome 19, analysis 3]
Statistical Analysis 10: Comparison: Placebo vs GSK249320 1 mg/kg; Placebo Vs GSK249320 1 mg/kg, Visit 7; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 3.04, 95% CI 2-sided [-5.53 to 11.61], Standard Error of Mean 4.205 — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 11: Comparison: Placebo vs GSK249320 5 mg/kg; Placebo Vs GSK249320 5 mg/kg, Visit 7; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = -2.58, 95% CI 2-sided [-11.5 to 6.32], Standard Error of Mean 4.376 — [estimate comment as in outcome 19, analysis 2]
Statistical Analysis 12: Comparison: Placebo vs GSK249320 15 mg/kg; Placebo Vs GSK249320 15 mg/kg, Visit 7; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 3.73, 95% CI 2-sided [-5.22 to 12.69], Standard Error of Mean 4.396 — [estimate comment as in outcome 19, analysis 3]

20. Secondary Outcome: Number of Participants With Modified Rankin Scale (mRS)
Description: The mRS was a 6 point scale that measured participant handicap by evaluating limitations in activity and changes in lifestyle. The mRS was staff-assessed and scored from 0=no symptoms at all, 1=no significant disability, 2=slight disability, 3=moderate disability, 4=moderate severe disability, 5=severe disability (severe disability, bedridden, incontinent and requiring constant nursing care and attention). The structured interview was used to administer the mRS. The mRS took approximately 15 minutes to complete when using the structured interview. Number of participants with mRS were reported as per the category of the score.
Time Frame: Day 30 and 90
Population: All subjects population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK249320 1 mg/kg | GSK249320 5 mg/kg | GSK249320 15 mg/kg
Number analyzed (Participants) | 17 | 8 | 9 | 8
Participants
  Visit 4 Day 30: number analyzed (Participants) | 14 | 8 | 9 | 7
  Visit 4 Day 30: mRS Score 0 | 0 | 0 | 0 | 0
  Visit 4 Day 30: mRS Score 1 | 2 | 2 | 1 | 2
  Visit 4 Day 30: mRS Score 2 | 3 | 1 | 3 | 0
  Visit 4 Day 30: mRS Score 3 | 3 | 3 | 3 | 3
  Visit 4 Day 30: mRS Score 4 | 4 | 2 | 2 | 2
  Visit 4 Day 30: mRS Score 5 | 2 | 0 | 0 | 0
  Visit 6 Day 90: number analyzed (Participants) | 14 | 8 | 8 | 6
  Visit 6 Day 90: mRS Score 0 | 0 | 1 | 1 | 0
  Visit 6 Day 90: mRS Score 1 | 3 | 1 | 2 | 2
  Visit 6 Day 90: mRS Score 2 | 5 | 2 | 2 | 1
  Visit 6 Day 90: mRS Score 3 | 3 | 4 | 2 | 0
  Visit 6 Day 90: mRS Score 4 | 3 | 0 | 1 | 2
  Visit 6 Day 90: mRS Score 5 | 0 | 0 | 0 | 1
Statistical Analysis 1: Comparison: Placebo vs GSK249320 1 mg/kg vs GSK249320 5 mg/kg vs GSK249320 15 mg/kg; Visit 4; Test type: Superiority or Other; p = 0.9260, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs GSK249320 1 mg/kg vs GSK249320 5 mg/kg vs GSK249320 15 mg/kg; Visit 6; Test type: Superiority or Other; p = 0.5647, Fisher Exact

21. Secondary Outcome: Change From Baseline of National Institutes of Health Stroke Scale (NIHSS)
Description: The NIHSS is a staff-assessed, 15 item, standardized, disease-specific, deficit scale which measures neurological impairment and is used to quantify participant status by measuring the severity of the stroke. The total NIHSS score ranged from 0 (No impairment) to 42 (severe impairment). Approximately 15 minutes were needed to complete the NIHSS. The NIHSS will be collected as part of the eligibility requirements to exclude participants who have a deficit that is either too mild or too severe. Only NIHSS certified study personnel recorded the NIHSS. Baseline assessments were recorded at Day 1 of the study. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. If either the Baseline or post-randomization value was missing, the change from Baseline was set to missing as well.
Time Frame: Baseline (Day 1), Day 10, 30 and 90
Population: All Subjects population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Placebo | GSK249320 1 mg/kg | GSK249320 5 mg/kg | GSK249320 15 mg/kg
Number analyzed (Participants) | 17 | 8 | 9 | 8
Score on scale
  Visit 3 Day 10: number analyzed (Participants) | 14 | 8 | 9 | 7
  Visit 3 Day 10 | -1.6 (1.79) | -3.1 (2.36) | -1.8 (1.72) | -4.4 (2.07)
  Visit 4 Day 30: number analyzed (Participants) | 14 | 8 | 9 | 7
  Visit 4 Day 30 | -3.7 (2.02) | -4.6 (2.13) | -4.0 (3.00) | -4.6 (2.23)
  Visit 6 Day 90: number analyzed (Participants) | 14 | 8 | 9 | 6
  Visit 6 Day 90 | -5.0 (2.91) | -6.3 (1.67) | -5.4 (2.77) | -2.7 (4.80)
Statistical Analysis 1: Comparison: Placebo vs GSK249320 1 mg/kg; Placebo Vs GSK249320 1 mg/kg, Visit 3; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Median Difference (Net) = -1.34, 95% CI 2-sided [-3.17 to 0.49], Standard Error of Mean 0.896 — Mean difference= GSK249320 1 mg/kg - Placebo Change from Baseline = Treatment + Visit + Treatment * Visit + Baseline
Statistical Analysis 2: Comparison: Placebo vs GSK249320 5 mg/kg; Placebo Vs GSK249320 5 mg/kg, Visit 3; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = -0.19, 95% CI 2-sided [-1.95 to 1.57], Standard Error of Mean 0.861 — Mean difference= GSK249320 5 mg/kg - Placebo Change from Baseline = Treatment + Visit + Treatment * Visit + Baseline
Statistical Analysis 3: Comparison: Placebo vs GSK249320 15 mg/kg; Placebo Vs GSK249320 15 mg/kg, Visit 3; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = -2.92, 95% CI 2-sided [-4.83 to -1.02], Standard Error of Mean 0.933 — Mean difference= GSK249320 15 mg/kg - Placebo Change from Baseline = Treatment + Visit + Treatment * Visit + Baseline
Statistical Analysis 4: Comparison: Placebo vs GSK249320 1 mg/kg; Placebo Vs GSK249320 1 mg/kg, Visit 4; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = -0.70, 95% CI 2-sided [-2.47 to 1.08], Standard Error of Mean 0.868 — Mean difference= GSK249320 1 mg/kg - Placebo Change from Baseline = Treatment + Visit + Treatment * Visit + Baseline
Statistical Analysis 5: Comparison: Placebo vs GSK249320 5 mg/kg; Placebo Vs GSK249320 5 mg/kg, Visit 4; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Median Difference (Net) = -0.27, 95% CI 2-sided [-1.98 to 1.44], Standard Error of Mean 0.834 — Mean difference= GSK249320 5 mg/kg - Placebo Change from Baseline = Treatment + Visit + Treatment * Visit + Baseline
Statistical Analysis 6: Comparison: Placebo vs GSK249320 15 mg/kg; Placebo Vs GSK249320 15 mg/kg, Visit 4; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Median Difference (Net) = -0.92, 95% CI 2-sided [-2.77 to 0.92], Standard Error of Mean 0.904 — Mean difference= GSK249320 15 mg/kg - Placebo Change from Baseline = Treatment + Visit + Treatment * Visit + Baseline
Statistical Analysis 7: Comparison: Placebo vs GSK249320 1 mg/kg; Placebo Vs GSK249320 1 mg/kg, Visit 6; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Median Difference (Net) = -1.03, 95% CI 2-sided [-3.64 to 1.57], Standard Error of Mean 1.278 — Mean difference= GSK249320 1 mg/kg - Placebo Change from Baseline = Treatment + Visit + Treatment * Visit + Baseline
Statistical Analysis 8: Comparison: Placebo vs GSK249320 5 mg/kg; Placebo Vs GSK249320 5 mg/kg, Visit 6; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = -0.37, 95% CI 2-sided [-2.97 to 2.24], Standard Error of Mean 1.278 — Mean difference= GSK249320 5 mg/kg - Placebo Change from Baseline = Treatment + Visit + Treatment * Visit + Baseline
Statistical Analysis 9: Comparison: Placebo vs GSK249320 15 mg/kg; Placebo Vs GSK249320 15 mg/kg, Visit 6; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Median Difference (Net) = -0.37, 95% CI 2-sided [-0.66 to 1.408], Standard Error of Mean 2.21 — Mean difference= GSK249320 15 mg/kg - Placebo Change from Baseline = Treatment + Visit + Treatment * Visit + Baseline

22. Secondary Outcome: Mean Barthel Total Score
Description: The Barthel was a staff-assessed, 10 item activities of daily living index that evaluated feeding, grooming, dressing, excretion (bowels, bladder and toilet skills), bathing, and mobility (transfers, walking, stairs). The total Barthel score ranged from either 0-20 or 0-100 depending on which scoring algorithm was used where 0= unable or dependent and 20 or 100= independent to perform daily activities. For this study, the 100 point scoring algorithm was used. The Barthel takes approximately 5-10 minutes to complete with the participant.
Time Frame: Day 30 and 90
Population: All subjects population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Placebo | GSK249320 1 mg/kg | GSK249320 5 mg/kg | GSK249320 15 mg/kg
Number analyzed (Participants) | 17 | 8 | 9 | 8
Score on scale
  Visit 4 Day 30: number analyzed (Participants) | 14 | 8 | 9 | 7
  Visit 4 Day 30 | 66.8 (36.19) | 86.3 (23.41) | 87.8 (20.63) | 78.6 (22.86)
  Visit 6 Day 90: number analyzed (Participants) | 14 | 8 | 8 | 6
  Visit 6 Day 90 | 81.8 (25.30) | 97.5 (3.78) | 92.5 (11.65) | 74.2 (29.40)
Statistical Analysis 1: Comparison: Placebo vs GSK249320 1 mg/kg; Placebo Vs GSK249320 1 mg/kg, Visit 4; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 19.46, 95% CI 2-sided [-6.11 to 45.04], Standard Error of Mean 12.584 — Mean difference= GSK249320 1 mg/kg - Placebo Barthel Total Score= Treatment + Visit + Treatment *Visit
Statistical Analysis 2: Comparison: Placebo vs GSK249320 5 mg/kg; Placebo Vs GSK249320 5 mg/kg, Visit 4; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 20.99, 95% CI 2-sided [-3.66 to 45.64], Standard Error of Mean 12.131 — Mean difference= GSK249320 5 mg/kg - Placebo Barthel Total Score= Treatment + Visit + Treatment *Visit
Statistical Analysis 3: Comparison: Placebo vs GSK249320 15 mg/kg; Placebo Vs GSK249320 15 mg/kg, Visit 4; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 11.79, 95% CI 2-sided [-14.9 to 38.50], Standard Error of Mean 13.143 — Mean difference= GSK249320 15 mg/kg - Placebo Barthel Total Score= Treatment + Visit + Treatment *Visit
Statistical Analysis 4: Comparison: Placebo vs GSK249320 1 mg/kg; Placebo Vs GSK249320 1 mg/kg, Visit 6; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 15.71, 95% CI 2-sided [-2.63 to 34.06], Standard Error of Mean 9.021 — Mean difference= GSK249320 1 mg/kg - Placebo Barthel Total Score= Treatment + Visit + Treatment *Visit
Statistical Analysis 5: Comparison: Placebo vs GSK249320 5 mg/kg; Placebo Vs GSK249320 5 mg/kg, Visit 6; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 11.56, 95% CI 2-sided [-6.38 to 29.50], Standard Error of Mean 8.835 — Mean difference= GSK249320 5 mg/kg - Placebo Barthel Total Score= Treatment + Visit + Treatment *Visit
Statistical Analysis 6: Comparison: Placebo vs GSK249320 15 mg/kg; Placebo Vs GSK249320 15 mg/kg, Visit 6; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = -7.49, 95% CI 2-sided [-27.1 to 12.08], Standard Error of Mean 9.641 — Mean difference= GSK249320 15 mg/kg - Placebo Barthel Total Score= Treatment + Visit + Treatment *Visit

23. Secondary Outcome: Mean Total Montreal Cognitive Assessment (MoCA) Score
Description: MoCA was an examiner-administered, screening instrument with good validity, reliability, sensitivity and specificity for mild cognitive dysfunction. The MoCA had been studied in stroke participants and was recommended as a tool to monitor and measure cognitive changes post stroke as part of the 2006 National Institute of Neurological Disorders and Stroke - Canadian Stroke Network Vascular Cognitive Impairment Harmonization Standards. The MoCA assesses eight cognitive domains of visuospatial skills, executive function, language, attention, concentration, working memory, memory, and orientation. Participants were asked to complete 14 activities which the examiner scored according to the standardized scoring instructions. While there was no set time limit imposed on a participant. The total MoCA score ranges from 0-30, where 0= worsening and 30 reflects normal cognitive function.
Time Frame: Day 5 and 90
Population: All Subjects population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Placebo | GSK249320 1 mg/kg | GSK249320 5 mg/kg | GSK249320 15 mg/kg
Number analyzed (Participants) | 17 | 8 | 9 | 8
Score on scale
  Visit 2 Day 5: number analyzed (Participants) | 14 | 8 | 9 | 8
  Visit 2 Day 5 | 19.4 (7.46) | 18.0 (9.94) | 15.2 (11.63) | 21.6 (9.30)
  Visit 6 Day 90: number analyzed (Participants) | 14 | 8 | 8 | 6
  Visit 6 Day 90 | 22.7 (5.27) | 21.6 (7.60) | 20.9 (8.72) | 22.8 (9.93)
Statistical Analysis 1: Comparison: Placebo vs GSK249320 1 mg/kg; Placebo Vs GSK249320 1 mg/kg, Visit 6; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = -0.34, 95% CI 2-sided [-4.12 to 3.43], Standard Error of Mean 1.849 — Mean difference= GSK249320 1 mg/kg - Placebo Day 90 MoCA = Treatment + Day 5 MoCA
Statistical Analysis 2: Comparison: Placebo vs GSK249320 5 mg/kg; Placebo Vs GSK249320 5 mg/kg, Visit 6; Test type: Superiority or Other; ANCOVA; Median Difference (Net) = -0.17, 95% CI 2-sided [-3.96 to 3.62], Standard Error of Mean 1.856 — Mean difference= GSK249320 5 mg/kg - Placebo Day 90 MoCA = Treatment + Day 5 MoCA
Statistical Analysis 3: Comparison: Placebo vs GSK249320 15 mg/kg; Placebo Vs GSK249320 15 mg/kg, Visit 6; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = -1.15, 95% CI 2-sided [-5.31 to 3.01], Standard Error of Mean 2.037 — Mean difference= GSK249320 15 mg/kg - Placebo Day 90 MoCA = Treatment + Day 5 MoCA

24. Secondary Outcome: Mean Geriatric Depression Scale (GDS)
Description: The short form GDS is a measure of depression developed specifically for use in elderly population and is sensitive and valid in the stroke population. The GDS was a participant-completed, 15 item questionnaire where each question referenced how the participant felt over the past week. Each question was answered with either a 'yes' or 'no' response. Of the 15 questions, 10 of them indicate depression when answered 'yes' (questions 2-4, 6, 8-10, 12, 14-15) and 5 indicate depression when answered 'no' (questions 1, 5, 7, 11, 13). Each question received a score of 1 point when the response was indicative of depression. Total score ranged from 0 to 15. the total score ranged from 0-15, where 0 implies no symptoms and higher score implies more severity of symptoms.
Time Frame: Day 5 and 90
Population: All Subjects population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Placebo | GSK249320 1 mg/kg | GSK249320 5 mg/kg | GSK249320 15 mg/kg
Number analyzed (Participants) | 17 | 8 | 9 | 8
Score on scale
  Visit 2 Day 5: number analyzed (Participants) | 14 | 8 | 8 | 8
  Visit 2 Day 5 | 4.5 (4.15) | 2.1 (1.36) | 5.1 (3.68) | 3.6 (2.67)
  Visit 6 Day 90: number analyzed (Participants) | 14 | 8 | 8 | 6
  Visit 6 Day 90 | 4.5 (3.48) | 2.8 (1.83) | 6.1 (3.91) | 3.8 (4.12)
Statistical Analysis 1: Comparison: Placebo vs GSK249320 1 mg/kg; Placebo Vs GSK249320 1 mg/kg, Visit 6; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = -0.24, 95% CI 2-sided [-3.12 to 2.63], Standard Error of Mean 1.408 — Mean difference= GSK249320 1 mg/kg - Placebo. Day 90 GDS Score= Treatment + Day 5 GDS Score
Statistical Analysis 2: Comparison: Placebo vs GSK249320 5 mg/kg; Placebo Vs GSK249320 5 mg/kg, Visit 6; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = 1.55, 95% CI 2-sided [-1.20 to 4.30], Standard Error of Mean 1.347 — Mean difference= GSK249320 5 mg/kg - Placebo Day 90 GDS Score= Treatment + Day 5 GDS Score
Statistical Analysis 3: Comparison: Placebo vs GSK249320 15 mg/kg; Placebo Vs GSK249320 15 mg/kg, Visit 6; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = -0.06, 95% CI 2-sided [-3.09 to 2.98], Standard Error of Mean 1.486 — Mean difference= GSK249320 15 mg/kg - Placebo. Day 90 GDS Score= Treatment+Day 5 GDS Score

25. Secondary Outcome: Mean Change in Transcranial Magnetic Stimulations (TMS) Evaluated by Peak to Peak MEP by % Stimulation Level
Description: TMS is an electrophysiological technique that was used to measure neurologic changes associated with recovery from stroke via alterations in the excitability of the motor system. Motor threshold measures reflect global excitability of the corticospinal pathway, including large pyramidal cells, excitatory/inhibitory interneurons, and spinal motorneurons. Motor threshold was recorded as the lowest stimulus intensity (in percent) eliciting motor evoked potentials (MEPs). Baseline assessments were recorded at Day 1 of the study. The change from Baseline was calculated by subtracting the Baseline values from the individual post -randomization values. If either the Baseline or post-randomization value was missing, the change from Baseline was set to missing as well.
Time Frame: Baseline (Day 1), Day 30 and 112
Population: All subjects population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change in stimulation
Arm/Group | Placebo | GSK249320 1 mg/kg | GSK249320 5 mg/kg | GSK249320 15 mg/kg
Number analyzed (Participants) | 17 | 8 | 9 | 8
Percent change in stimulation
  Stimulation Level 100%, Visit 4 Day 30: number analyzed (Participants) | 10 | 5 | 6 | 3
  Stimulation Level 100%, Visit 4 Day 30 | 0.289 (0.6046) | -0.068 (0.4125) | -1.560 (3.9411) | 0.030 (0.1600)
  Stimulation Level 100%, Visit 7 Day 112: number analyzed (Participants) | 9 | 5 | 5 | 2
  Stimulation Level 100%, Visit 7 Day 112 | -0.021 (0.1365) | 0.116 (0.5811) | 0.148 (0.3270) | 0.465 (0.6293)
  Stimulation Level 110%, Visit 4 Day 30: number analyzed (Participants) | 10 | 5 | 6 | 3
  Stimulation Level 110%, Visit 4 Day 30 | 0.525 (0.9065) | 1.420 (2.5622) | -1.535 (4.3653) | 0.283 (0.6950)
  Stimulation Level 110%, Visit 7 Day 112: number analyzed (Participants) | 9 | 5 | 5 | 2
  Stimulation Level 110%, Visit 7 Day 112 | 0.168 (0.4176) | 0.690 (1.0786) | 0.298 (0.5837) | 1.850 (2.5032)
  Stimulation Level 120%, Visit 4 Day 30: number analyzed (Participants) | 10 | 4 | 6 | 3
  Stimulation Level 120%, Visit 4 Day 30 | 0.741 (1.3249) | 2.023 (1.8115) | -0.557 (4.9402) | 0.640 (1.3393)
  Stimulation Level 120%, Visit 7 Day 112: number analyzed (Participants) | 9 | 5 | 5 | 2
  Stimulation Level 120%, Visit 7 Day 112 | 0.590 (1.5803) | 0.728 (0.4908) | 0.490 (0.4887) | 3.035 (4.0093)
  Stimulation Level 130%, Visit 4 Day 30: number analyzed (Participants) | 10 | 4 | 6 | 3
  Stimulation Level 130%, Visit 4 Day 30 | 0.802 (1.6584) | 1.180 (0.6988) | -0.697 (4.9586) | 0.697 (1.6763)
  Stimulation Level 130%, Visit 7 Day 112: number analyzed (Participants) | 9 | 4 | 5 | 2
  Stimulation Level 130%, Visit 7 Day 112 | 0.636 (1.8215) | 0.100 (1.0296) | 0.706 (0.6750) | 3.335 (4.4760)
  Stimulation Level 140%, Visit 4 Day 30: number analyzed (Participants) | 10 | 4 | 6 | 3
  Stimulation Level 140%, Visit 4 Day 30 | 1.042 (1.8231) | 1.100 (1.5979) | -0.768 (4.6784) | 0.867 (2.7265)
  Stimulation Level 140%, Visit 7 Day 112: number analyzed (Participants) | 9 | 4 | 5 | 2
  Stimulation Level 140%, Visit 7 Day 112 | 0.742 (2.1058) | -0.050 (1.6503) | 0.954 (1.1362) | 3.040 (4.0447)
Statistical Analysis 1: Comparison: Placebo vs GSK249320 1 mg/kg; Stimulation Level 100%, Visit 4 Day 30; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Median Difference (Net) = -0.289, 95% CI 2-sided [-0.841 to 0.264], Standard Error of Mean 0.2639 — Mean difference= GSK249320 1 mg/kg - Placebo Change from Baseline= Treatment + Visit + Treatment* Visit + Baseline
Statistical Analysis 2: Comparison: Placebo vs GSK249320 5 mg/kg; Stimulation Level 100%, Visit 4 Day 30; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = -0.310, 95% CI 2-sided [-0.862 to 0.241], Standard Error of Mean 0.2637 — Mean difference= GSK249320 5 mg/kg - Placebo Change from Baseline= Treatment + Visit + Treatment* Visit + Baseline
Statistical Analysis 3: Comparison: Placebo vs GSK249320 15 mg/kg; Stimulation Level 100%, Visit 4 Day 30; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Median Difference (Net) = -0.303, 95% CI 2-sided [-0.966 to 0.361], Standard Error of Mean 0.3172 — Mean difference= GSK249320 15 mg/kg - Placebo Change from Baseline= Treatment + Visit + Treatment* Visit + Baseline
Statistical Analysis 4: Comparison: Placebo vs GSK249320 1 mg/kg; Stimulation Level 100%, Visit 7 Day 112; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Median Difference (Net) = 0.204, 95% CI 2-sided [-0.184 to 0.593], Standard Error of Mean 0.1841 — Mean difference= GSK249320 1 mg/kg - Placebo Change from Baseline= Treatment + Visit + Treatment* Visit + Baseline
Statistical Analysis 5: Comparison: Placebo vs GSK249320 5 mg/kg; Stimulation Level 100%, Visit 7 Day 112; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 0.105, 95% CI 2-sided [-0.284 to 0.494], Standard Error of Mean 0.1846 — Mean difference= GSK249320 5 mg/kg - Placebo Change from Baseline= Treatment + Visit + Treatment* Visit + Baseline
Statistical Analysis 6: Comparison: Placebo vs GSK249320 15 mg/kg; Stimulation Level 100%, Visit 7 Day 112; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 0.416, 95% CI 2-sided [-0.132 to 0.965], Standard Error of Mean 0.2602 — Mean difference= GSK249320 15 mg/kg - Placebo Change from Baseline= Treatment + Visit + Treatment* Visit + Baseline
Statistical Analysis 7: Comparison: Placebo vs GSK249320 1 mg/kg; Stimulation Level 110%, Visit 4 Day 30; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 1.156, 95% CI 2-sided [-0.650 to 2.961], Standard Error of Mean 0.8652 — Mean difference= GSK249320 1 mg/kg - Placebo Change from Baseline= Treatment + Visit + Treatment* Visit + Baseline
Statistical Analysis 8: Comparison: Placebo vs GSK249320 5 mg/kg; Stimulation Level 110%, Visit 4 Day 30; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = -0.518, 95% CI 2-sided [-2.249 to 1.213], Standard Error of Mean 0.8324 — Mean difference= GSK249320 5 mg/kg - Placebo Change from Baseline= Treatment + Visit + Treatment* Visit + Baseline
Statistical Analysis 9: Comparison: Placebo vs GSK249320 15 mg/kg; Stimulation Level 110%, Visit 4 Day 30; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = -0.269, 95% CI 2-sided [-2.436 to 1.898], Standard Error of Mean 1.0383 — Mean difference= GSK249320 15 mg/kg - Placebo Change from Baseline= Treatment + Visit + Treatment* Visit + Baseline
Statistical Analysis 10: Comparison: Placebo vs GSK249320 1 mg/kg; Stimulation Level 110%, Visit 7 Day 112; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 0.806, 95% CI 2-sided [-0.420 to 2.031], Standard Error of Mean 0.5862 — Mean difference= GSK249320 1 mg/kg - Placebo Change from Baseline= Treatment + Visit + Treatment* Visit + Baseline
Statistical Analysis 11: Comparison: Placebo vs GSK249320 5 mg/kg; Stimulation Level 110%, Visit 7 Day 112; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = -0.007, 95% CI 2-sided [-1.183 to 1.168], Standard Error of Mean 0.5640 — Mean difference= GSK249320 5 mg/kg - Placebo Change from Baseline= Treatment + Visit + Treatment* Visit
Statistical Analysis 12: Comparison: Placebo vs GSK249320 15 mg/kg; Stimulation Level 110%, Visit 7 Day 112; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 1.506, 95% CI 2-sided [-0.064 to 3.077], Standard Error of Mean 0.7570 — Mean difference= GSK249320 15 mg/kg - Placebo Change from Baseline= Treatment + Visit + Treatment* Visit + Baseline
Statistical Analysis 13: Comparison: Placebo vs GSK249320 1 mg/kg; Stimulation Level 120%, Visit 4 Day 30; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 1.644, 95% CI 2-sided [-1.056 to 4.344], Standard Error of Mean 1.2976 — Mean difference= GSK249320 1 mg/kg - Placebo Change from Baseline= Treatment + Visit + Treatment* Visit + Baseline
Statistical Analysis 14: Comparison: Placebo vs GSK249320 5 mg/kg; Stimulation Level 120%, Visit 4 Day 30; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = -0.231, 95% CI 2-sided [-2.681 to 2.219], Standard Error of Mean 1.1762 — Mean difference= GSK249320 5 mg/kg - Placebo Change from Baseline= Treatment + Visit + Treatment* Visit + Baseline
Statistical Analysis 15: Comparison: Placebo vs GSK249320 15 mg/kg; Stimulation Level 120%, Visit 4 Day 30; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = -0.184, 95% CI 2-sided [-3.279 to 2.910], Standard Error of Mean 1.4796 — Mean difference= GSK249320 15 mg/kg - Placebo Change from Baseline= Treatment + Visit + Treatment* Visit + Baseline
Statistical Analysis 16: Comparison: Placebo vs GSK249320 1 mg/kg; Stimulation Level 120%, Visit 7 Day 112; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 0.622, 95% CI 2-sided [-1.428 to 2.672], Standard Error of Mean 0.9746 — Mean difference= GSK249320 1 mg/kg - Placebo Change from Baseline= Treatment + Visit + Treatment* Visit + Baseline
Statistical Analysis 17: Comparison: Placebo vs GSK249320 5 mg/kg; Stimulation Level 120%, Visit 7 Day 112; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = -0.602, 95% CI 2-sided [-2.560 to 1.356], Standard Error of Mean 0.9340 — Mean difference= GSK249320 5 mg/kg - Placebo Change from Baseline= Treatment + Visit + Treatment* Visit + Baseline
Statistical Analysis 18: Comparison: Placebo vs GSK249320 15 mg/kg; Stimulation Level 120%, Visit 7 Day 112; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 2.063, 95% CI 2-sided [-0.610 to 4.736], Standard Error of Mean 1.2810 — Mean difference= GSK249320 15 mg/kg - Placebo Change from Baseline= Treatment + Visit + Treatment* Visit + Baseline
Statistical Analysis 19: Comparison: Placebo vs GSK249320 1 mg/kg; Stimulation Level 130%, Visit 4 Day 30; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 1.556, 95% CI 2-sided [-1.494 to 4.607], Standard Error of Mean 1.4588 — Mean difference= GSK249320 1 mg/kg - Placebo Change from Baseline= Treatment + Visit + Treatment* Visit + Baseline
Statistical Analysis 20: Comparison: Placebo vs GSK249320 5 mg/kg; Stimulation Level 130%, Visit 4 Day 30; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = -0.531, 95% CI 2-sided [-3.102 to 2.041], Standard Error of Mean 1.2336 — Mean difference= GSK249320 5 mg/kg - Placebo Change from Baseline= Treatment + Visit + Treatment* Visit + Baseline
Statistical Analysis 21: Comparison: Placebo vs GSK249320 15 mg/kg; Stimulation Level 130%, Visit 4 Day 30; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = -0.185, 95% CI 2-sided [-3.471 to 3.101], Standard Error of Mean 1.5697 — Mean difference= GSK249320 15 mg/kg - Placebo Change from Baseline= Treatment + Visit + Treatment* Visit + Baseline
Statistical Analysis 22: Comparison: Placebo vs GSK249320 1 mg/kg; Stimulation Level 130%, Visit 7 Day 112; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 0.686, 95% CI 2-sided [-1.996 to 3.367], Standard Error of Mean 1.2689 — Mean difference= GSK249320 1 mg/kg - Placebo Change from Baseline= Treatment + Visit + Treatment* Visit + Baseline
Statistical Analysis 23: Comparison: Placebo vs GSK249320 5 mg/kg; Stimulation Level 130%, Visit 7 Day 112; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = -0.556, 95% CI 2-sided [-2.838 to 1.726], Standard Error of Mean 1.0822 — Mean difference= GSK249320 5 mg/kg - Placebo Change from Baseline= Treatment + Visit + Treatment* Visit + Baseline
Statistical Analysis 24: Comparison: Placebo vs GSK249320 15 mg/kg; Stimulation Level 130%, Visit 7 Day 112; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 2.219, 95% CI 2-sided [-0.884 to 5.322], Standard Error of Mean 1.4792 — Mean difference= GSK249320 15 mg/kg - Placebo Change from Baseline= Treatment + Visit + Treatment* Visit + Baseline
Statistical Analysis 25: Comparison: Placebo vs GSK249320 1 mg/kg; Stimulation Level 140%, Visit 4 Day 30; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 1.631, 95% CI 2-sided [-1.696 to 4.958], Standard Error of Mean 1.5890 — Mean difference= GSK249320 1 mg/kg - Placebo Change from Baseline= Treatment + Visit + Treatment* Visit + Baseline
Statistical Analysis 26: Comparison: Placebo vs GSK249320 5 mg/kg; Stimulation Level 140%, Visit 4 Day 30; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = -0.508, 95% CI 2-sided [-3.219 to 2.203], Standard Error of Mean 1.2985 — Mean difference= GSK249320 5 mg/kg - Placebo Change from Baseline= Treatment + Visit + Treatment* Visit + Baseline
Statistical Analysis 27: Comparison: Placebo vs GSK249320 15 mg/kg; Stimulation Level 140%, Visit 4 Day 30; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 0.110, 95% CI 2-sided [-3.369 to 3.588], Standard Error of Mean 1.6603 — Mean difference= GSK249320 15 mg/kg - Placebo Change from Baseline= Treatment + Visit + Treatment* Visit + Baseline
Statistical Analysis 28: Comparison: Placebo vs GSK249320 1 mg/kg; Stimulation Level 140%, Visit 7 Day 112; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 0.852, 95% CI 2-sided [-2.446 to 4.150], Standard Error of Mean 1.5675 — Mean difference= GSK249320 1 mg/kg - Placebo Change from Baseline= Treatment + Visit + Treatment* Visit + Baseline
Statistical Analysis 29: Comparison: Placebo vs GSK249320 5 mg/kg; Stimulation Level 140%, Visit 7 Day 112; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = -0.357, 95% CI 2-sided [-3.074 to 2.359], Standard Error of Mean 1.2918 — Mean difference= GSK249320 5 mg/kg - Placebo Change from Baseline= Treatment + Visit + Treatment* Visit + Baseline
Statistical Analysis 30: Comparison: Placebo vs GSK249320 15 mg/kg; Stimulation Level 140%, Visit 7 Day 112; Test type: Superiority or Other; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 1.686, 95% CI 2-sided [-1.937 to 5.308], Standard Error of Mean 1.7306 — Mean difference= GSK249320 15 mg/kg - Placebo Change from Baseline= Treatment + Visit + Treatment* Visit + Baseline

26. Secondary Outcome: Serum Levels of the S100β Protein
Description: The serum sample for S100β collected on Day 1 (predose, 1, 6, 12 and 24 hour) and Day 5 and was analyzed for levels. Serum levels of S100β protein were recorded as log transformed values therefore the negative values are reported.
Time Frame: Day 1 (Pre-dose, Post dose 1, 6, 24 hour), Day 5
Population: All Subjects population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: log (ug per liter)
Arm/Group | Placebo | GSK249320 1 mg/kg | GSK249320 5 mg/kg | GSK249320 15 mg/kg
Number analyzed (Participants) | 17 | 8 | 9 | 8
log (ug per liter)
  Visit 1, Day 1- Pre-dose: number analyzed (Participants) | 13 | 4 | 8 | 8
  Visit 1, Day 1- Pre-dose | -1.021 (1.3655) | -1.224 (1.0676) | -0.978 (1.3218) | -1.624 (1.1256)
  Visit 1, Day 1- 1 hour post-dose: number analyzed (Participants) | 13 | 4 | 8 | 8
  Visit 1, Day 1- 1 hour post-dose | -1.024 (1.2038) | -0.785 (1.3917) | -1.130 (1.4363) | -1.615 (1.2312)
  Visit 1, Day 1 - 6 hour post-dose: number analyzed (Participants) | 13 | 4 | 8 | 8
  Visit 1, Day 1 - 6 hour post-dose | -0.851 (1.4014) | -1.251 (1.0449) | -0.895 (1.4683) | -1.135 (0.7006)
  Visit 1, Day 1 - 24 hour post-dose: number analyzed (Participants) | 13 | 4 | 8 | 7
  Visit 1, Day 1 - 24 hour post-dose | -1.053 (1.4309) | -1.329 (0.9649) | -0.744 (1.3523) | -1.644 (1.0244)
  Visit 2, Day 5: number analyzed (Participants) | 9 | 3 | 8 | 8
  Visit 2, Day 5 | -1.050 (1.0039) | -1.697 (0.7264) | -0.920 (1.1960) | -1.821 (0.9974)

ADVERSE EVENTS:
Time Frame: AEs were collected up to Day 112
Description: All subject population was used to report AEs.
Arm/Group | Placebo | GSK249320 1 mg/kg | GSK249320 5 mg/kg | GSK249320 15 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/8 | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 3/17 | 1/8 | 3/9 | 3/8
Other Adverse Events (participants affected / at risk) | 9/17 | 6/8 | 7/9 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=17) | GSK249320 1 mg/kg (N=8) | GSK249320 5 mg/kg (N=9) | GSK249320 15 mg/kg (N=8)
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Helicobacter infection (Infections and infestations) | 0 | 0 | 1 | 0
Peridiverticulitis (Infections and infestations) | 0 | 0 | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=17) | GSK249320 1 mg/kg (N=8) | GSK249320 5 mg/kg (N=9) | GSK249320 15 mg/kg (N=8)
Constipation (Gastrointestinal disorders) | 2 | 2 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1
Clostridial infection (Infections and infestations) | 0 | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 1 | 1
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 2 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 1
Protein total abnormal (Investigations) | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.